

# PM1183-B-003-11

# A Multicenter Phase II Clinical Trial of PM01183 in BRCA 1/2-Associated or Unselected Metastatic Breast Cancer

STATISTICAL ANALYSIS PLAN

NCT Code: 01525589

Version: 3.0

Date: 10-December-2018

# **TABLE OF CONTENTS**

| 1 | TZ | UDY RATIONALE | 6 |
|---|---|---|---|
| 2 | | UDY DESIGN | 7 |
| 3 | | JECTIVES AND ENDPOINTS | |
| , | 3.1 | Primary Objective | 8 |
| | 3.2 | Secondary Objectives | 8 |
| | 3.3 | Endpoints | 8 |
| 4 | | ΓΙΕΝΤS EVALUABILITY CRITERIA | 9 |
| • | 4.1 | Included Population | 9 |
| | | Efficacy Populations | 9 |
| | 4.3 | Safety Population | 10 |
| 5 | | MPLE CONSIDERATIONS | 10 |
| ٠ | 5.1 | Sample Size | 10 |
| 6 | | ATISTICAL METHODOLOGY FOR EFFICACY | 10 |
| - | 6.1 | Planned Analysis and Definitions | 10 |
| | 6.2 | Efficacy Analysis Methods | 11 |
| | 6.2 | 1 Primary Endpoint | 12 |
| | | 2 Secondary Endpoints | 12 |
| 7 | STA | ATISTICAL METHODOLOGY FOR SAFETY | 13 |
| | 7.1 | 1 Toxicity and Adverse Events | 13 |
| | 7.2 | Clinical Laboratory Evaluation | 13 |
| | 7.3 | Vital Signs, Physical Examination, Left Ventricular Ejection Fraction and | |
| | Electr | ocardiogram Findings | 14 |
| | 7.4 | Deaths and Other Serious Adverse Events | 14 |
| 8 | OT | HER ANALYSIS | 14 |
| | 8.1 | Patient Disposition and Treatment/Study Discontinuation | 14 |
| | 8.2 | Protocol Deviations | 14 |
| | 8.3 | Baseline and Demographic Data | 14 |
| | 8.4 | Treatment Administration | 15 |
| | 8.5 | Subsequent Therapy | 16 |
| | 8.6 | Pharmacokinetic Analysis | 16 |
| | 8.7 | Pharmacogenomic Analysis | 16 |
| | 8.8 | Imputation of Incomplete Dates | 16 |
| | 8.9 | Subgroup Analysis | 17 |
| | 8.10 | Methods for Handling Missing Data | 17 |
| | 8.11 | Interim and Group Sequential Analysis | 17 |
| | 8.12 | Identification of Fixed or Random Effects Models | 18 |
| 9 | | ATISTICAL SOFTWARE | 18 |
| | | NDIX I | 19 |
| 1( | | dy Patients | 19 |
| | 10.1 | Patient Disposition | 19 |
| | 10.2 | Reasons for Treatment Discontinuation | 20 |
| | 10.3 | Protocol Deviations | 22 |
| 1 | l Eff | icacy Evaluation | 23 |

| 11 | 1.1 | Demographic and Other Baseline Characteristics | 23 |
|---|---|---|---|
| | 11.1.1 | Patient Characteristics at Baseline | 23 |
| | 11.1.2 | Disease at Diagnosis and Current Disease | 23 |
| | | Prior History | 25 |
| | 11.1.4 | Prior Anticancer Therapy | 25 |
| | 11.1.5 | Physical Examination and Performance Status at Baseline | 26 |
| | | Vital Signs, Electrocardiogram, LVEF and other tests. | 27 |
| | 11.1.7 | Hematological Values at Baseline | 28 |
| | 11.1.8 | Biochemical Values at Baseline | 29 |
| | 11.1.9 | Coagulation Values at Baseline | 30 |
| | 11.1.10 | Signs and Symptoms at Baseline | 30 |
| | 11.1.11 | Concomitant Therapy and Procedures at Baseline | 31 |
| 11 | 1.2 | Measurements of Treatment Compliance | 34 |
| 11 | 1.3 | Efficacy Analysis | 35 |
| | 11.3.1 | Primary Analysis | 35 |
| | 11.3.2 | Secondary Analysis | 36 |
| | 11.3.3 | Exploratory Multivariate Analysis | 39 |
| 12 | Safety A | analysis | 41 |
| 12.1 | | Extent of Exposure | 41 |
| 12 | 2.1.1 | Treatment Administration | 41 |
| | 12.1.2 | Cycle Delays | 41 |
| | 12.1.3 | Dose Reductions | 43 |
| | 12.1.4 | Infusions Temporarily Interrupted | 45 |
| | 12.1.5 | Prophylactic Medication Administration | 45 |
| 12 | | Adverse Events | 45 |
| | 12.2.1 | Adverse Events | 45 |
| | 12.2.2 | Display of Adverse Events | 46 |
| | 12.2.3 | Evolution of signs and symptoms during the treatment | 48 |
| 12 | 2.3 | Serious Adverse Events and Deaths. | 48 |
| | 12.3.1 | Serious Adverse Events | 48 |
| | 12.3.2 | Deaths | 49 |
| 12 | 2.4 | Clinical Laboratory Evaluation | 49 |
| | 12.4.1 | Hematological Abnormalities | 50 |
| | 12.4.2 | Biochemical Abnormalities | 50 |
| | 12.4.3 | Coagulation Abnormalities | 52 |
| | 12.4.4 | Laboratory Values Over Time | 53 |
| 12 | 2.5 | Physical Findings, PS, LVEF, ECG and Other Tests Related to Safety | 64 |
| | | Physical Findings and PS (ECOG) | 64 |
| | | LVEF, ECG and Other Related Tests | 64 |
| | 2.6 | Concomitant Therapy / Procedures According to the ATC Classification. | 65 |
| 13 | DB Listi | <del>-</del> | 67 |
| 14 | SAP Ve | rsion History | 68 |

# ABBREVIATIONS AND GLOSSARY

| ADDKEVIA | HONS AND GLOSSARY |
|---|---|
| AE(s) | Adverse Event(s) |
| ALT | Alanine Aminotransferase |
| AP | Alkaline Phosphatase |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BL | Baseline |
| BRCA1/2 | Breast Cancer 1 or Breast Cancer 2 Susceptibility Gene |
| BSA | Body Surface Area |
| C | Cycle |
| CI | Confidence Interval |
| СРК | Creatine Phosphokinase |
| CR | Complete Response |
| CRF | Case Report Form |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DB | Database |
| DR | Duration of Response |
| DNA | Deoxyribonucleic Acid |
| ECG | Electrocardiogram |
| ЕСНО | Echocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| FD | Flat Dose |
| G-CSF | Granulocyte-Colony Stimulating Factor |
| GGT | Gamma-glutamyltransferase |
| HER-2 | Human Epidermal Growth Factor Receptor 2 |
| IB | Investigator's Brochure |
| i.v. | Intravenous(ly) |
| K | Potassium |
| LDH | Lactate Dehydrogenase |
| LVEF | Left Ventricular Ejection Fraction |
| MBC | Metastatic Breast Cancer |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MUGA | Multiple-gated Acquisition Scan |
| NA | Sodium / Not applicable |
| NCI | National Cancer Institute |
| NCI-CTC | National Cancer Institute Common Toxicity Criteria |
| NCI-CTCAE | National Cancer Institute Common Terminology Criteria for Adverse Events |

| NE | Not Evaluable |
|--------|----------------------------------------------|
| NOS | Not Otherwise Specified |
| ORR | Overall Response Rate |
| os | Overall Survival |
| PARPi | Poly ADP Ribose Polymerase inhibitor |
| PD | Progressive Disease |
| PFS | Progression-free Survival |
| PGx | Pharmacogenomics |
| PK/PD | Pharmacokinetics/Pharmacodynamic |
| PR | Partial Response |
| PS | Performance Status |
| PT | Prothrombin Time/Preferred Term |
| PTT | Partial Thromboplastin Time |
| q3wk | Every Three Weeks |
| RD | Recommended Dose |
| RECIST | Response Evaluation Criteria In Solid Tumors |
| SAE(s) | Serious Adverse Event(s) |
| SD | Stable Disease |
| SOC | System Organ Class |
| ULN | Upper Limit of Normal |
| UK | Unknown |
| vs. | Versus |
| WBC | White Blood Cells |
| WHO | World Health Organization |
| Wk(s) | Week(s) |
| y | Year |

### 1 STUDY RATIONALE

Metastatic breast cancer (MBC) is a clinically heterogeneous and an aggressive disease from which most patients will ultimately die. Unfortunately a cure by the means of currently available treatment options still seems an elusive goal. Cytotoxic chemotherapy remains a crucial component of the therapeutic armamentarium and there is a need to develop more selective approaches to identify subgroups of patients with higher tumor sensitivity that may benefit the most.

PM01183 is a new chemical entity that induces double-strand DNA breaks through binding to the DNA minor groove. Results of the COMPARE analysis (see protocol reference 20) revealed that is unlikely that this drug shares a similar mechanism of action with any of the other 98 standard cytotoxic agents compared.

PM01183 has significant *in vitro* and *in vivo* wide antitumor activity, particularly in several breast cancer models.

PM01183 exposure primarily induces DNA damage, particularly to homologous recombinant deficient cells *in vitro* (see IB); thus, patients with BRCA deleterious mutation might be more sensitive to its antitumor effects than other patients. In order to test this hypothesis, two Cohorts of patients with advanced breast cancer will be prospectively evaluated in the trial according to their germline BRCA1/2 mutation status: known mutation (BRCA+, Cohort A) vs. unselected (BRCA- or -UK, Cohort B).

The goal of the trial is, on one hand, to find out whether the presence of a BRCA 1/2 mutation in Cohort A is associated with a higher response rate in MBC patients; and, on the other hand, to explore and benchmark the activity of PM01183 in MBC unselected patients. The study design has taken into account the higher sample heterogeneity of Cohort B by planning the recruitment of more patients in this group. Also, according to the BRCA status in the trial setting, a response rate of 40% or more in Cohort A (sample of patients with known deleterious BRCA 1/2 mutations) will be considered clinically worthy of further research, as well as a response rate of 25% or more in Cohort B.

The first-in-human phase I clinical trial found a RD of 7.0 mg FD of PM01183 when given as a one-hour i.v. infusion q3wk. This dose was safe, tolerable and manageable for a highly selected patient population. In particular, PM01183 induced predictable and short-lasting non-febrile neutropenia as the most relevant toxicity (up to 40% of patients treated at the RD). None of the patients treated at the RD were older than 75 years and/or had PS >1. Therefore, it is uncertain at this time if PM01183 RD is as tolerable and safe for a particularly vulnerable and frail population given the degree of myelosuppresion observed so far. Because toxicity, especially in aging patients, is usually an important consideration in order to select the more suitable treatment, it seems safer to exclude patients over 75 years old and/or with PS≥2 until more information regarding safety and pharmacokinetics of the drug becomes available.

#### 2 STUDY DESIGN

This is a multicenter, open-label, exploratory, phase II clinical trial evaluating the efficacy and safety of PM01183 administration to patients with previously treated MBC, as follows.

Two Cohorts of MBC patients will be prospectively evaluated in the trial according to germline BRCA1/2 status (mutated [Cohort A] vs. unselected [Cohort B]). A third Cohort (Cohort A1) will include advanced breast cancer patients with deleterious BRCA1/2 mutation status who received prior treatment with poly (ADP-ribose) polymerase (PARP) inhibitors:

- <u>Cohort A (BRCA+ Cohort)</u>: At least 53 evaluable patients with previously known deleterious BRCA1/2 mutation status at study entry.
- <u>Cohort A1 (BRCA+/PARPi Cohort):</u> 20 evaluable patients with known deleterious BRCA1/2 mutation status and prior treatment with PARP inhibitors (PARPi).
- <u>Cohort B (unselected Cohort)</u>: At least 64 evaluable patients without known deleterious BRCA1/2 mutation status at study entry, i.e., either:
  - o Patients known to have no deleterious BRCA1/2 mutations (BRCA-), or
  - Patients whose BRCA 1/2 mutation status is unknown (BRCA-UK); BRCA1/2 germline mutation status will be assessed in PM01183 responding patients in this subgroup.

In patients included in Cohort B who respond to PM01183 treatment and whose BRCA 1/2 mutation status is unknown at study entry, an analysis will be performed in order to confirm or exclude deleterious germline BRCA 1/2 mutation. To this end, a blood sample will be collected at the time of response. If a BRCA 1/2 mutation is found in her sample then the patient will be analyzed along with patients included in Cohort A.

The primary efficacy endpoint of the study is the overall response rate (ORR), defined as the percentage of patients with a response, either complete (CR) or partial (PR), according to RECIST v1.1 (protocol section 8.1).

An interim analysis based on the primary endpoint (ORR) is planned after 20 and 30 evaluable patients have been treated in Cohorts A and B, respectively (see protocol section 8.2 for details). No interim analysis is planned for Cohort A1. If less than four out of 20 patients in Cohort A, or less than three out of 30 patients in Cohort B achieve an objective confirmed response, recruitment to that Cohort will be terminated. Otherwise, recruitment will continue until at least 53 and 64 evaluable patients are included in Cohort A and Cohort B, respectively. Sample size and Cohort design will be re-evaluated at this point in order to estimate the 95% confidence interval (CI) with the desired precision. Recruitment to either Cohort (e.g., Cohort B) might be halted while interim analysis is being performed, if appropriate.

Patients will receive treatment in the absence of progressive disease (PD) or unacceptable toxicity for as long as it is considered to be in their own benefit (see protocol section 6.2.1.2 for details).

Patients will be evaluated using clinical and laboratory assessments before each treatment cycle (protocol sections 6.3 and 6.6). Appropriate radiological and/or clinical tumor

assessments will be done every six weeks until evidence of PD (protocol section 7.1). Patients no longer receiving study treatment will be followed up for survival (protocol section 6.8).

Any treatment-related AE will be followed until recovery to grade  $\leq 1$  or stabilization of symptoms, whenever possible (protocol section 7.2). Reasons for dose reduction, treatment delays and/or treatment discontinuation will be documented as appropriate.

### 3 OBJECTIVES AND ENDPOINTS

### 3.1 Primary Objective

• To assess the antitumor activity of PM01183 in terms of ORR, according to RECIST v1.1, in each Cohort of MBC patients.

### 3.2 Secondary Objectives

- To further characterize the antitumor activity of PM01183 in terms of duration of response (DR), clinical benefit [ORR or stable disease lasting over three months (SD > 3 months)], PFS, and one-year overall survival (1y-OS).
- To evaluate whether the presence of a known germline mutation in BRCA1/2 predicts response to PM01183 in MBC patients.
- To explore the activity of PM01183 in specific breast cancer subpopulations according to hormonal receptor status, HER-2 overexpression, number and/or type of prior therapies, or according to other available histological/molecular classifications.
- To evaluate the safety profile of this PM01183 administration schedule (Day 1, q3wk) in this patient population.
- To analyze the pharmacokinetics (PK) of PM01183 in this patient population.
- To explore PK/PD (pharmacokinetic / pharmacodynamic) correlations, if applicable.
- To evaluate the pharmacogenomic (PGx) expression profile of selected putative markers potentially predictive of response to PM01183, in tissues from archived tumor samples.

### 3.3 Endpoints

#### Primary endpoint:

 Overall response rate (ORR) in the population evaluable for efficacy, according to RECIST v1.1.

### Secondary endpoints:

• Duration of response (DR).

- Clinical benefit, defined as the percentage of patients with ORR or SD > 3 months, according to RECIST v1.1.
- Progression-free survival (PFS).
- Overall survival rate at one year (1y-OS).
- Treatment safety: AEs, serious AEs (SAEs) and laboratory abnormalities will be graded according to the NCI-CTCAE (v4).
- PK analysis and PK/PD correlation, if applicable.
- PGx expression profile, in tissues from archived tumor samples.

#### 4 PATIENTS EVALUABILITY CRITERIA

The study population will include patients with MBC histologically proven.

Analysis sets definitions:

- "All Included Patients" analysis set is defined as all patients recorded in the database who are included in the trial, independently of whether they have received the study drug or not.
- ° "All Treated Patients" analysis set is defined as all included patients who have received at least part of one infusion of PM01183.
- "All Evaluable Patients" analysis set is defined as all eligible patients who have at least one complete infusion of PM01183, and either have at least one assessment (as per RECIST v1.1) or have been categorized as "treatment failures". Patients who discontinue treatment due to any treatment-related toxicity before an appropriate tumor assessment has been performed or those withdrawn after more than two weeks on treatment without any formal evaluation will be defined as "treatment failures". These patients will be included as inevaluable for response in the analysis of objective response as per RECIST v1.1, although they will not need to be replaced as they will be considered evaluable for efficacy.
- ° "All Responder Patients" analysis set is defined as all evaluable patients who have had CR or PR as overall best response according to the RECIST v1.1 criteria.

#### 4.1 Included Population

The "All Included Patients" data set will be used for the descriptive analysis of baseline characteristics.

### 4.2 Efficacy Populations

The "All Evaluable Patients" analysis set will be used for the primary endpoint analysis of ORR and for the secondary endpoints of PFS, 1y-OS and clinical benefit rate.

The "All Responder Patients" set will be used for the secondary endpoint analysis of DR.

### 4.3 Safety Population

The safety analysis for the secondary endpoint will be based on the "All Treated Patients" analysis set.

### 5 SAMPLE CONSIDERATIONS

#### 5.1 Sample Size

The primary endpoint for this phase II study is to evaluate ORR.

### • Cohort A (BRCA+):

At least 53 evaluable patients will be recruited to test the null hypothesis that ORR is 20% or less (p  $\leq$  0.20) vs. the alternative hypothesis that 40% or more patients have objective response (p  $\geq$  0.4). With these assumptions, if the number of evaluable patients with objective response is  $\geq$  17, then this would allow the rejection of the null hypothesis.

### Cohort A1 (BRCA+/PARPi):

At least 20 evaluable patients will be recruited for an exploratory analysis: if the number of patients responding is  $\geq 4$  (20%), the lower limit of the exact binomial 95% confidence interval will be higher than 5% and thus lack of activity in this subpopulation will be ruled out.

### • Cohort B (unselected):

At least 64 evaluable patients will be recruited to test the null hypothesis that ORR is 10% or less (p  $\leq$  0.10) vs. the alternative hypothesis that 25% or more patients have objective response (p  $\geq$  0.25). With these assumptions, if the number of evaluable patients with objective response is  $\geq$  12, then this would allow the rejection of the null hypothesis.

The variance of the standardized tests is based on the null hypothesis. The type I error (alpha) associated with this one-sided test is 0.025 and the type II error (beta) is <0.1; hence, statistical power is > 90%.

Futility analysis controlled by the Gamma family boundary will be performed when 20 and 30 patients have been evaluated in Cohorts A [Gm(-2)] and B [Gm(-1.5)], respectively. If less than four out of 20 patients in Cohort A, or less than three patients out of 30 in Cohort B achieve an objective response, recruitment to that Cohort will be stopped. About 110 evaluable patients are finally expected to be included in the three Cohorts: Cohort A (BRCA+), Cohort A1 (BRCA+/PARPi), and Cohort B (unselected).

#### 6 STATISTICAL METHODOLOGY FOR EFFICACY

Frequency tables will be performed for categorical variables, whereas continuous variables will be described by means of summary tables that will include the median, minimum, and maximum of each variable.

### 6.1 Planned Analysis and Definitions

Primary endpoint

The primary study analysis will be based on the ORR in the "All Evaluable Patients" analysis set.

*Overall response rate (ORR)* is calculated as the number of patients who have had CR or PR as overall best response according to the RECIST v1.1 criteria, divided by the number of patients in the "All Evaluable Patients" analysis set.

#### Secondary endpoint

The following time-related parameters would be analyzed according to available follow-up data:

**Duration of response (DR)** is defined as time from first observation of response to the date of disease progression, recurrence of death. Other causes will be censored. Although the responses have to be confirmed according to RECIST v1.1 criteria, the first documentation, not the confirmation, will be taken into account to calculate DR. Patients who progress or die will be considered to have had an event, except if this event occurs after the start of subsequent antitumor therapy, in which case the patient will be censored at the time of last disease assessment prior to or on the first day of the first subsequent antitumor therapy.

Clinical benefit rate is calculated as the number of patients who have had CR or PR or SD  $\geq$  3 months as overall best response according to the RECIST v1.1 criteria, divided by the number of patients in the "All Evaluable Patients" analysis set.

**Progression-free survival (PFS)** is defined as the time from start of treatment to the date of documented progressive disease (PD) by RECIST v1.1 criteria or death (regardless of the cause of death), whichever comes first. Patients who progress or die will be considered to have had an event, except if this event occurs after the start of subsequent antitumor therapy, in which case the patient will be censored at the time of last disease assessment prior to or on the first day of the first subsequent antitumor therapy. If the patient is lost for the assessment of progression during the follow-up period, or has more than one missing follow-up between the date of last tumor assessment and the date of progression, death or further antitumor therapy, the PFS will be censored at the date of last valid disease assessment before the missing evaluations.

Overall survival (OS) is defined as the time from the date of start of treatment to the date of death or last contact. 1 year overall survival (1y-OS) is defined as the Kaplan-Meier estimate of the probability of patients alive after 12 months from the date of start of treatment.

### 6.2 Efficacy Analysis Methods

Continuous variables will be tabulated by Cohort and presented with summary statistics (i.e., median and range). Categorical variables will be summarized by Cohort in frequency tables by means of counts and percentages.

### 6.2.1 Primary Endpoint

Exact binomial estimates with 95% confidence intervals (CIs) will be calculated for the analysis of the main endpoint (ORR according to RECIST v1.1 criteria).

#### 6.2.2 Secondary Endpoints

Time-to-event endpoints (DR, PFS and OS) and their set time estimates (i.e. PFS3, PFS6 and 1y-OS) will be analyzed according to the Kaplan-Meier method.

A log-rank test or Cox regression for time-to-event endpoints could be performed as supportive analysis to compare both Cohorts.

If relevant, efficacy parameters versus baseline covariates will be analyzed and appropriate test will be used (i.e., the Fisher exact test and logistic regression for categorical variables, the log-rank test or Cox regression for time-to-event variables, etc.).

If appropriate, exploratory multivariate models (main effects or including interaction terms, if appropriate) will include all prognostic factors/covariates widely reported and recognized by oncologists: Cohort (BRCA (+) vs. BRCA (-) or unknown), BRCA (1 vs. 2 in cohorts A and A1), initial dose (7 mg FD vs 3.5 mg/m<sup>2</sup>), age, age at diagnosis, race (Caucasian vs. other), baseline Eastern Cooperative Oncology Group performance status (ECOG PS) (0 vs. >0), histology type (Ductal vs. lobular carcinoma), histology grade (poorly vs. other), stage at diagnosis, primary tumor site (unilateral breast vs. bilateral), hormone receptor positive (estrogen or progesterone receptor +, or both +) vs. triple negative, HER-2 receptor (positive vs. negative), site of current disease such as liver metastases (yes vs. no), CNS metastases (yes vs. no), lung metastases (yes vs. no), non-visceral (including bone, skin, subcutaneous and lymph node vs. other), number of prior metastatic sites (1 vs. >1), body mass index (BMI), height, weight, body surface area (BSA), time from diagnosis to first infusion, prior surgery (yes vs. no), prior radiotherapy (yes vs. no), prior advanced treatment lines, prior advanced chemotherapy lines (0-1 vs. 2-3), prior anthracyclines (ves vs. no), prior taxane (yes vs. no), prior platinum (yes vs. no), prior PARPi (yes vs. no), last prior therapy PFS, first advanced chemotherapy PFS, last advanced chemotherapy PFS, PFS for anthracycline, taxane and platinum therapy, hormonotherapy (yes vs no), adjuvant/neoadjuvant therapy (yes vs no), platinum-free interval (in months), presence of any bulky (< 50 mm vs. ≥ 50 mm) lesion, albumin at baseline, CA-15.3 or 27.29 at baseline, any relevant concomitant medication at baseline (to be determinate by the oncologist) (yes vs. no) and the sum of all target lesion diameters.

All variables with a good percentage of valid cases (approximately  $\geq$  90%) and with a p-value lower than 0.10 in the univariate analysis will be included in the exploratory multivariate analysis. Within the multivariate stepwise Logistic/Cox regression analysis, the chosen significance level for entering an explanatory variable into the model will be 0.05 (for all variables not in the model, the one with the smallest p-value is entered if the p-value is less than or equal to the specified significance level). The significance level for removing an explanatory variable from the model is 0.05 (for all variables in the model, the one with the largest p-value will be removed if the p-value exceeds the specified significance level). The parameter estimates, hazard ratios and p-values for hazard ratios of the variables retained in the model will be presented.

If appropriate, multivariate analysis will be produced for a relevant subgroup of patients (e.g. by cohort).

### 7 STATISTICAL METHODOLOGY FOR SAFETY

The safety analysis for the secondary endpoints will be based on the "All Treated Patients" analysis set.

Patients will be evaluable for safety if they received at least one partial or complete infusion of PM01183

# 7.1.1 Toxicity and Adverse Events

All the adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

The toxicity evaluation will be coded with the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 4.

As far as all the toxicities are concerned, the NCI-CTCAE grade will be used wherever an NCI-CTCAE grading exists. Otherwise, the severity will be noted. As a convention, the term «Grade» will always be used. Toxicities will be described according to the worst NCI-CTCAE grade or, for toxicities which do not form the subject of NCI-CTCAE classification, according to the worst severity.

Summary of overall AEs will be done by System Organ Class (SOC) and Preferred Term (PT), by severity (worst toxicity grade), by relationship to the study drug and by AE outcome. Tables will be sorted by SOC/PT coded with MedDRA.

A frequency table will be made for the AEs leading to cycle delay, dose reduction or withdrawal of study medication. Adverse events with outcome of death will also be presented by relationship to the study drugs.

### 7.2 Clinical Laboratory Evaluation

Laboratory results will be classified according to the NCI-CTCAE version 4.

The following hematological values (worst grade per patient and per cycle during treatment) will be displayed: white blood cells (WBC) count, neutrophil count, lymphocyte count, platelet count and hemoglobin.

Overall cross tabulation will be presented for the worst grade during treatment versus the baseline toxicity grading of anemia, lymphopenia, neutropenia, leukopenia and thrombocytopenia.

If a grade 3-4 neutropenia or thrombocytopenia increase occur during a cycle of treatment, the first day it reached the onset value (counting from the start of the cycle) and the duration of the abnormality (until recovery to grade  $\leq 2$ ), will be tabulated.

Similarly, the following biochemical values (worst grade per patient and per cycle during treatment) will be displayed: alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, alkaline phosphatase (AP), creatine phosphokinase (CPK),

creatinine, gamma-glutamyltransferase (GGT), calcium (corrected by albumin levels), potassium (K), sodium (NA), magnesium, glucose, phosphorus, triglycerides and albumin.

If a grade 3-4 AST or ALT increase occur during a cycle of treatment, both the day it peaked (counting from the start of the cycle) and the duration of the abnormality (until recovery to grade  $\leq 2$ ), will be tabulated.

Overall cross tabulation will be presented for the worst grade during treatment versus the baseline toxicity grading of biochemical abnormalities.

# 7.3 Vital Signs, Physical Examination, Left Ventricular Ejection Fraction and Electrocardiogram Findings

Tabulation will be made summarizing the performance status, body weight, left ventricular ejection fraction (LVEF) and electrocardiogram (ECG) abnormalities at baseline and during the treatment, if appropriate, for each patient.

#### 7.4 Deaths and Other Serious Adverse Events

Deaths and other SAEs will be tabulated.

#### 8 OTHER ANALYSIS

Continuous variables will be tabulated and presented with summary statistics (i.e., median and range).

Categorical variables will be summarized in frequency tables by means of counts and percentages. Percentages in the summary tables will be rounded and may therefore not always add up to exactly 100%.

### 8.1 Patient Disposition and Treatment/Study Discontinuation

The number of patients included in the study, the number of patients treated and the number of patients evaluable for the main endpoint, will be shown. Also, accrual by center and country and the main dates of the study will be displayed. Reasons for treatment discontinuation and for study discontinuation will be tabulated.

#### 8.2 Protocol Deviations

Analysis of inclusion/exclusion criteria deviations, retreatment restrictions, concomitant medication and clinically relevant discontinuations, among others, will be done as described in Appendix I.

### 8.3 Baseline and Demographic Data

Baseline data such as demographics, cancer history, prior therapy, prior relevant history, signs and symptoms, electrocardiogram, LVEF, physical examination, vital signs, laboratory values and concomitant medication, coded according to the Word Health Organization (WHO) Anatomical Therapeutic Chemical (ATC) classification system, will be described following standard tables detailed in Appendix I.

Age, baseline weight, height, and body surface area (BSA) will be summarized descriptively.

Age will be calculated based on the date of birth and the date of informed consent.

Baseline weight and height are recorded on the CRF.

Baseline BSA will be calculated using the Dubois & Dubois formula:

$$BSA(m^2) = 0.007184 \times weight(kg)^{0.425} \times height(cm)^{0.725}$$

Age categories and race will be summarized with frequency counts.

Baseline Eastern Cooperative Oncology Group (ECOG) performance status (PS) will be summarized with frequency counts.

For the cancer history: time from initial diagnosis, time from metastatic disease and time from last progression before the study entry will be summarized. This time calculations will be shown in months and summarized descriptively. Histology and characteristics of the current disease will be tabulated.

Previous relevant medical history (other than cancer) will be listed.

A frequency tabulation of the number of patients with and the different types of previous surgery, radiotherapy, or therapy (number of lines) will be given.

Signs and symptoms at baseline will be displayed by tabulation of frequencies according to NCI-CTCAE version 4 toxicity grades. Signs and symptoms will be listed.

In case of pre-treatment characteristics with multiple measurements per subject before the start of treatment (laboratory assessments, vital signs) the baseline measurement will be considered the last value prior to or on the first day of treatment.

Baseline and demography characteristics in different subgroups of analysis (i.e. cohorts) will be compared by means of Fisher's exact test (categorical variables) and Mann-Whitney-Wilcoxon (continuous variables).

#### 8.4 Treatment Administration

Total cumulative dose, dose intensity and relative dose intensity, time on treatment, cycle delays and dose reductions will be described following standard tables detailed in Appendix I

Total cumulative dose, expressed in mg, is the sum of all the study drug doses from the first cycle until last cycle, including the dose received in last cycle.

Patients will be considered to be on-treatment for the duration of their treatment and 30 days following the last treatment dose. If the patient starts any new antitumor therapy outside this clinical trial or dies within 30 days of last treatment dose, the date of administration of this new therapy or the date of death will be considered the date of treatment discontinuation.

However, as a convention, the duration of the last cycle is considered to be 21 days (instead of 30 days) for dose intensity calculation purposes.

Intended dose intensity (mg/m²) is the planned dose per cycle divided by the planned number of weeks per cycle.

Absolute dose intensity (mg) is the actual cumulative dose divided by the number of weeks of treatment. Relative dose intensity (%) is the ratio of absolute dose intensity divided by the intended dose intensity.

The item of the case report form (CRF) «Infusion delayed: yes/no» will be used to calculate the delayed cycles. For those cycles considered as delayed by the investigator, the delay will be calculated as:

Delay: Date of current drug administration – Date of previous drug administration – 21.

The infusion of the first cycle will be excluded from all calculations regarding cycle delays and modifications.

### 8.5 Subsequent Therapy

A table summarizing the subsequent therapies received after treatment discontinuation will be shown.

#### 8.6 Pharmacokinetic Analysis

This analysis will be detailed in a separate document.

# 8.7 Pharmacogenomic Analysis

This analysis will be detailed in a separate document.

# 8.8 Imputation of Incomplete Dates

The dates of certain historical or current clinical activities are key component for statistical analysis. An incomplete date results from a missing day, month or year; in that case, the missing figure can be imputed allowing for the calculation of variables, such duration and time to certain event. However, when all of them, day, month and year, are missing no imputation will be done.

#### Before registration

If the day of a month is unknown, then the imputed day will be the 15<sup>th</sup> of the month; if the month is also unknown, then the imputed date will be the 1<sup>st</sup> of July. This assumption will only be valid if the imputed date occurs earlier than the first dose administration date; otherwise the imputed date will be the first day of the first dose administration month date (i.e. 01/ first dose administration month date/year).

### Between treatment start and end of treatment

All date variables during treatment where information is needed and is not fully available, for example adverse events or concomitant medications, will be subject of imputation by means of SAS programming. If the day of a date is unknown then the imputed day will be 1, if the month and/or year is also unknown then the imputed date will 1/January (this assumption will be valid if the imputed date is not earlier than the treatment start date; otherwise, the imputed date will be the treatment start date).

### After end of treatment

To ensure the most conservative approach for the time-to-event variables (i.e., DR, PFS and OS), which can be affected by missing values, the following rules will be implemented: if the day of a date is unknown then the imputed day will be the 1<sup>st</sup>; if the month is also unknown, then the imputed date will be the 1<sup>st</sup> of July. This assumption will be valid if the imputed date occurs later than the last drug administration date; otherwise the imputed date will be the date of the last drug administration plus the predefined cycle length (i.e., 21 days if PM01183), except if the patient dies before, in which case the date of death minus 1 will be used.

### 8.9 Subgroup Analysis

The analysis will be done by Cohort and additionally, if clinically appropriate, the Cohorts might be pooled into one, whenever differences between Cohorts are considered not relevant. In such case, the point estimates and their 95% CIs will be also reassessed in order to obtain more accurate calculations.

Efficacy subgroup analysis will be performed in Cohort A according to prior treatment with platinum (Yes vs. No), BRCA status (BRCA1 vs. BRCA2), hormonal status (Triple negative vs. HR+), number of advanced chemotherapy lines, prior PARPi (Yes vs. No)and starting dose (7 mg FD vs. 3.5 mg/m²).

Additional efficacy subgroup analysis will be performed in Cohorts A+A1 according to prior PARPi (Yes vs. No). Safety subgroup analysis will be performed according to starting dose (7 mg FD vs. 3.5 mg/m²), these analysis include laboratory abnormalities and adverse events.

If clinically relevant, other subgroup analysis may be performed in order to explore the activity of PM01183 in specific breast cancer subpopulations.

No differentiation by center is planned.

#### 8.10 Methods for Handling Missing Data

Missing values will be tabulated with their frequency but they will not be included in the calculation of percentages.

### 8.11 Interim and Group Sequential Analysis

An interim analysis based on the primary endpoint (ORR) is planned after 20 and 30 evaluable patients have been treated in Cohorts A and B, respectively. If less than four out of 20 patients in Cohort A, or less than three out of 30 patients in Cohort B achieve an objective confirmed response (CR or PR according to RECIST v1.1), recruitment to that Cohort will be terminated. Otherwise, recruitment will continue until at least 53 and 64 evaluable patients are included in Cohort A and Cohort B, respectively. Sample size and Cohort design will be re-evaluated at this point in order to estimate the 95% confidence interval (CI) with the desired precision. For further analysis details, see section 5.1 Sample size.

# 8.12 Identification of Fixed or Random Effects Models

Not applicable

# 9 STATISTICAL SOFTWARE

Medidata Rave® EDC will be used for data entry and clinical data management.

EAST v.5.4 has been used to calculate sample size. SAS version 9 will be used for all statistical analysis outputs.

### APPENDIX I

Every output will be displayed by Cohort and/or total and they will be clearly identified with a label. To maintain simplicity, nested categories are not presented.

# 10 Study Patients

### 10.1 Patient Disposition

Main characteristics concerning inclusion in the study, withdrawal from the study and protocol deviations will be displayed in this section.

Table 10.1.1 Number of patients included, treated and evaluable for the main endpoint.

| | N | % |
|---------------------------------|---|---|
| Included patients | | |
| Eligible patients* | | |
| Treated patients | | |
| Evaluable patients for efficacy | | |

<sup>(\*)</sup>Patients meeting all inclusion criteria and not meeting any exclusion criteria.

Listing 10.1.2 Patients who do not meet all the inclusion criteria.

| Patient id. | Criteria number(s) and description |
|---|---|
| Listing 10.1.3 Pat | ients who meet any exclusion criteria. |
| Patient id. Criteria number(s) and description | |
| Listing 10.1.4 No | n-evaluable patients for efficacy analysis. |
| Patient id. | Reason |

| Listing 10.1 | 5 Non-evaluable natients for safety (Non-treat | ed natients) |
|--------------|------------------------------------------------|--------------|

| Elbumg 10.1.0 11 | on evaluable patients for safety (1 ton treated patients). |
|---|---|
| Patient id. | Reason |

Table 10.1.6 Patients accrual by institution

| | | | N | % |
|--------------------------|-----------|---------------|---|---|
| | Country 1 | Institution 1 | | |
| | | Total | | |
| | | Institution 1 | | |
| No. of patients included | | | | |
| | | Total | | |
| | | Institution 1 | | |
| | Total | | | |
| | | Total | | |
| | Country 1 | Institution 1 | | |
| | | Total | | |
| | | Institution 1 | | |
| No. of patients treated | | | | |
| | | Total | | |
| | | Institution 1 | | |
| | Total | ••• | | |
| | | Total | | |

# Table 10.1.7 Study dates

| | Total |
|-----------------------------------------|-------|
| Date of first registration | |
| Date of first dose of the first patient | |
| Date of last registration | |
| Date of first dose of the last patient | |
| Date of last dose | |
| Date of last follow-up* | |

<sup>(\*)</sup> Last follow-up, exam or procedure before clinical cut-off or study closure

# 10.2 Reasons for Treatment Discontinuation

Table 10.2.1 Treatment discontinuation

| Reason | N | % |
|-------------------------------------|---|---|
| Progressive disease | | |
| Treatment related adverse event | | |
| Non Treatment related adverse event | | |
| Patient refusal to treatment | | |
| Death (due to toxicity)* | | |
| Death (non-treatment-related)** | | |
| Investigator's decision*** | | |
| Other *** | | |
| Total | | |

<sup>(\*)</sup> Cause of death = Study drug related Adverse Event; (\*\*) Cause of death = Malignant disease, Non-study drug related AE or Other; (\*\*\*) See Listing 10.2.2

Listing 10.2.2 Reasons for treatment discontinuation other than progressive disease.

| Patient id. | Reason | Last cycle | Comments |
|-------------|--------|------------|----------|

Table 10.2.3 Reasons for treatment discontinuation by cycles received

| Reason | Last cycle | | | |
|-------------------------------------|------------|---|-----|-------|
| | 1 | 2 | ••• | Total |
| Progressive disease | | | | |
| Treatment related adverse event | | | | |
| Non Treatment related adverse event | | | | |
| Patient refusal to treatment | | | | |
| Death (due to toxicity)* | | | | |
| Death (non-treatment-related)** | | | | |
| Investigator's decision*** | | | | |
| Other *** | | | | |
| Total | | | | |

<sup>(\*)</sup> Cause of death = Study drug related Adverse Event; (\*\*) Cause of death = Malignant disease, Non study drug related AE or Other; (\*\*\*) See Listing 10.2.2

When the reason for discontinuation is a study treatment-related adverse event or study treatment-related death, identify patients and describe them in depth here.

Listing 10.2.4 Treatment discontinuation due to AEs

| Patient id. | Last<br>Cycle | Preferred term code | Adverse event reported (verbatim) | Grade | Relationship | Onset<br>date | Resolved<br>date | Seriousness criteria |
|---|---|---|---|---|---|---|---|---|

### Table 10.2.5 Study discontinuation

| Reason | N | % |
|--------------------------------------|---|---|
| Never treated* | | |
| Study termination (clinical cut-off) | | |
| Patient's follow-up completed | | |
| Patient's refusal | | |
| Death (due to toxicity)** | | |
| Death (non-treatment-related)*** | | |
| Lost to follow-up | | |
| Other **** | | |
| Total | | |

<sup>(\*)</sup> See Listing 10.2.6; (\*\*) Cause of death = Study drug related Adverse Event; (\*\*\*) Cause of death = Malignant disease, Non study drug related AE or Other; (\*\*\*\*) Specify (see listing 10.2.7)

#### Listing 10.2.6 Patients included but not treated

| Patient id. | Off-study reason |
|-------------|------------------|

Listing 10.2.7 Study discontinuation due to other reason

| Patient id. | Specify |
|-------------|---------|

# 10.3 Protocol Deviations

Listing 10.3.1 Protocol deviations

| Patient id. | Deviation type | Description |
|-------------|----------------|-------------|

# 11 Efficacy Evaluation

# 11.1 Demographic and Other Baseline Characteristics

### 11.1.1 Patient Characteristics at Baseline

Table 11.1.1.1 Baseline characteristics: Age at treatment registration

| | N | Median | Min | Max |
|-------------|---|--------|-----|-----|
| Age (years) | | | | |

Table 11.1.1.2 Baseline characteristics: Age grouped

| | N | % |
|-------|---|------|
| 18-XX | X | XX.X |
| XX-YY | | |
| ≥65 | | |
| Total | | |

#### Table 11.1.1.3 Baseline characteristics: Race

| | N | % |
|-----------|---|------|
| Caucasian | X | XX.X |
| Asian | | |
| Black | | |
| Other* | | |
| Total | | |

<sup>(\*)</sup> See Listing 11.1.1.4;

Listing 11.1.1.4 Other race, specify

| Patient id. | Specify |
|-------------|---------|

# 11.1.2 Disease at Diagnosis and Current Disease

Table 11.1.2.1 Time from first diagnosis to registration

| | N | Median | Min | Max |
|--------------------------------------|---|--------|-----|-----|
| Time from diagnosis to randomization | | | | |
| (months) | | | | |

### Table 11.1.2.2 Site of disease at diagnosis

| | N | % |
|--------------|---|------|
| Right breast | X | XX.X |
| Left breast | | |
| Bilateral | | |
| Total | | |

# Table 11.1.2.3 Histology type at diagnosis

| | N | % |
|-------------------|---|------|
| Ductal Carcinoma | X | XX.X |
| Lobular Carcinoma | | |
| Total | | |

Table 11.1.2.4 Histology grade at diagnosis

| | N | % |
|---------------------------|---|------|
| Well differentiated | X | XX.X |
| Moderately differentiated | | |
| Poorly differentiated | | |
| Unknown | | |
| Total | | |

# Table 11.1.2.5 Stage at diagnosis

| | N | % |
|-------|---|------|
| | X | XX.X |
| Total | | |

# Table 11.1.2.6 BRCA in Arm A and Arm A1 (deletereous mutation).

| | N | % |
|--------|---|------|
| BRCA 1 | X | XX.X |
| BRCA 2 | | |
| Both | | |

### Table 11.1.2.7 BRCA in Arm B.

| | N | % |
|----------|---|------|
| Negative | X | XX.X |
| Unknown | | |

# Table 11.1.2.8 Receptor status. Current disease.

| | Positive % | | Negative | |
|-----------------------|------------|------|----------|------|
| | | | N | % |
| Estrogen receptor | X | XX.X | X | XX.X |
| Progesterone receptor | | | | |
| HER-2 Receptor | | | | |

### Table 11.1.2.9 Hormonal status

| | N | % |
|---------------------------------------|---|------|
| Triple negative | X | XX.X |
| ER and/or PR positive + HER2 negative | | |
| ER and/or PR positive + HER2 positive | | |
| ER and PR negative + HER2 positive | | |
| Total | | |

# Table 11.1.2.10 Time from Metastatic disease to registration

| | N | Median | Min | Max |
|---------------------------------------|---|--------|-----|-----|
| Time from metastatic disease (months) | | | | |

# Table 11.1.2.11 Time from last progression before the study entry

| | N | Median | Min | Max |
|---------------------------|---|--------|-----|-----|
| Time from last PD (weeks) | | | | |

Table 11.1.2.12 Sites of metastatic disease. Current disease.

| | N | % |
|------------|---|------|
| Lymph node | X | XX.X |
| Bone | | |
| Lung | | |
| Liver | | |
| Pleura | | |

# Table 11.1.2.13 Number of sites at baseline

| No. of sites | N | % |
|----------------|---|------|
| 1 | X | XX.X |
| 2 | | |
| Total | | |
| Median (Range) | | |

# 11.1.3 Prior History

# Table 11.1.3.1 Prior history

| SOC | Preferred Term | N | % |
|----------------------------|----------------|---|---|
| Gastrointestinal disorders | Constipation | | |
| | Diarrhea NOS | | |
| | ••• | | |

Listing 11.1.3.2 Prior history (Ongoing events)

| Patient id. | Description (Literal) | SOC | PT | Onset date |
|-------------|-----------------------|-----|----|------------|

# 11.1.4 Prior Anticancer Therapy

# Table 11.1.4.1 Patients with prior sugery

| Prior surgery | N | % |
|---------------|---|-----|
| Yes | X | X.X |
| No | | |
| Total | | |

# Table 11.1.4.2 Patients with prior radiotherapy

| Prior radiotherapy | N | % |
|--------------------|---|-----|
| Yes | X | X.X |
| No | | |
| Total | | |

Table 11.1.4.3 Number of lines of prior therapy

| No. of systemic lines | N | % |
|----------------------------------------|---|------|
| 1 | X | XX.X |
| Total | | |
| Median (Range) | | |
| Setting | N | % |
| Adjuvant | X | XX.X |
| Neoadjuvant | | |
| Both | | |
| Advanced | | |
| No. of advanced chemotherapy lines | N | % |
| 1 | X | XX.X |
| Total | | |
| Median (Range) | | |
| Prior chemotherapy regimens | N | % |
| Anthracycline and taxane | X | XX.X |
| Anthracycline, taxane and capecitabine | | |
| Platinum | | |
| No. of hormone* therapy lines | N | % |
| 1 | X | XX.X |
| Total | | |
| Median (Range) | | |

<sup>(\*)</sup> Hormone therapy will be identified by the oncologist;

# Table 11.1.4.4 Prior anticancer agents

| Antineoplastic and immunomodulating agents (ATC-class.) | N | % |
|---------------------------------------------------------|---|------|
| Antineoplastic agents (L01) | X | XX.X |
| Alkylating agents | | |
| Nitrogen mustard analogues | | |
| Alkyl sulphonates | | |

# 11.1.5 Physical Examination and Performance Status at Baseline

Table 11.1.5.1 Baseline physical examination

| | N | % |
|----------|---|-----|
| Normal | X | X.X |
| Abnormal | | |
| Total | | |

Table 11.1.5.2 Baseline physical examination: BSA, Weight and Height

| | N | Median | Min | Max |
|-----------------------|---|--------|-----|-----|
| BSA (m <sup>2</sup> ) | | | | |
| Weight (Kg) | X | X.X | X.X | X.X |
| Height (cm) | | | | |

Table 11.1.5.3 Baseline characteristics: ECOG Performance Status

| PS (ECOG) | N | % |
|-----------|---|------|
| 0 | X | XX.X |
| 1 | | |
| 2 | | |
| Total | | |

### 11.1.6 Vital Signs, Electrocardiogram, LVEF and other tests.

For vital signs, electrocardiogram, LVEF and other tests, the last examination available before treatment will be described in the following tables.

Table 11.1.6.1 Baseline characteristics: Vital signs

| Parameter | N | Median | Min | Max |
|---------------------------------|---|--------|-----|-----|
| Heart rate (beats/min) | | | | |
| Systolic blood pressure (mmHg) | | | | |
| Diastolic blood pressure (mmHg) | | | | |
| Temperature (°C) | | | | |

Table 11.1.6.2 Baseline characteristics: Electrocardiogram result

| ECG | N | % |
|-----------|---|------|
| Normal | X | XX.X |
| Abnormal* | | |
| Total | | |

<sup>(\*)</sup>See listing 11.1.6.4 for details

Table 11.1.6.3 Baseline characteristics: Electrocardiogram values

| Parameter | N | Median | Min | Max |
|--------------------|---|--------|-----|-----|
| PR interval (msec) | | | | |
| Heart rate (bpm) | | | | |
| QT interval (msec) | | | | |
| QRS complex (msec) | | | | |
| QTc Fridericia | | | | |

Listing 11.1.6.4 Patients with abnormal electrocardiogram

| Patien id. | Abnormality | Details* | Reason for<br>clinically<br>indicated<br>repeat | PR interval (msec) | Heart rate (bpm) | QT interval (msec) | QRS<br>complex<br>(msec) | QTc<br>Fridericia |
|---|---|---|---|---|---|---|---|---|

<sup>(\*)</sup>For non-significant abnormalities, for further details see prior medical history or Signs and symptoms

Table 11.1.6.5 Baseline characteristics: Left Ventricular Ejection Fraction (LVEF)

| LVEF | N | % |
|-----------|---|------|
| Normal | X | XX.X |
| Abnormal* | | |
| Total | | |

<sup>(\*)</sup>See listing 11.1.6.7 for details

Table 11.1.6.6 Baseline characteristics: LVEF values.

| LVEF (%) by Method | N | Median | Min | Max |
|--------------------|---|--------|-----|-----|
| ЕСНО | | | | |
| MUGA | | | | |
| Both | | | | |

### Listing 11.1.6.7 Patients with abnormal LVEF

| Patient id. | Abnormality | Details* | Reason for clinically indicated repeat | Method | LVEF (%) | Institution normal range |
|---|---|---|---|---|---|---|

<sup>(\*)</sup>For non-significant abnormalities, for further details see prior medical history or Signs and symptoms;

Table 11.1.6.8 Baseline characteristics: Pregnancy test

| Pregnancy test | N | % |
|----------------|---|------|
| Positive | X | XX.X |
| Negative | | |
| NA* | | |
| Total | | |

<sup>(\*)</sup> Specify reasons

Table 11.1.6.9 Baseline characteristics: Adequate contraception

| | 1 1 | |
|------------------------|-----|------|
| Adequate birth control | N | % |
| Yes | X | XX.X |
| No | | |
| NA* | | |
| Total | | |

<sup>(\*)</sup> Specify reasons

# 11.1.7 Hematological Values at Baseline

Table 11.1.7.1 Hematological abnormalities at baseline

| | N | Gr | ade<br>1 | <br>Gr | ade<br>4 | Al | 1* |
|------------------|---|----|----------|--------|----------|----|----|
| | | N | % | <br>N | % | N | % |
| Leukopenia | | | | | | | |
| Anemia | | | | | | | |
| Thrombocytopenia | | | | | | | |
| Neutropenia | | | | | | | |
| Lymphopenia | | | | | | | |

<sup>(\*)</sup>Any grade

Table 11.1.7.2 Hematology values at baseline

| | N | Median | Min | Max |
|----------------------------------|---|--------|-----|-----|
| Hemoglobin (g/dL) | | | | |
| Platelets (10 <sup>9</sup> /L) | | | | |
| WBC $(10^9/L)$ | | | | |
| Neutrophils (10 <sup>9</sup> /L) | | | | |
| Lymphocytes (10 <sup>9</sup> /L) | | | | |
| Monocytes (10 <sup>9</sup> /L) | | | | |

Listing 11.1.7.3 Hematological tests not assessed at baseline

| 8 | |
|-------------|-----------|
| Patient id. | Lab. test |

Listing 11.1.7.4 Hematological abnormalities at baseline. Grade  $\geq 2$ 

| Patient id | Parameter | Value | Units | Grade |
|------------|-----------|-------|-------|-------|

### 11.1.8 Biochemical Values at Baseline

Table 11.1.8.1 Biochemical abnormalities at baseline

| | N | Gr | ade<br>1 | <br>Gr | ade<br>4 | Al | 1* |
|--------------------------|---|----|----------|--------|----------|----|----|
| | | N | % | <br>N | % | N | % |
| AST increased | | | | | | | |
| ALT increased | | | | | | | |
| Total bilirubin increase | | | | | | | |
| AP increased | | | | | | | |
| ••• | | | | | | | |
| Hyperglycemia | | | | | | | |
| Hypoglycemia | | | | | | | |

<sup>(\*)</sup>Any grade

Table 11.1.8.2 Biochemical values at baseline

| | N | Median | Min | Max |
|-------------------------|---|--------|-----|-----|
| AST (xULN) | | | | |
| ALT (IU/L) | | | | |
| Direct bilirubin (xULN) | | | | |
| Total bilirubin (xULN) | | | | |
| AP (xULN) | | | | |
| LDH (xULN) | | | | |
| CPK (xULN) | | | | |
| GGT (xULN) | | | | |
| Creatinine (xULN) | | | | |
| Troponin T (ng/mL) | | | | |

Listing 11.1.8.3 Biochemical tests not assessed at baseline

| Patient id. | Lab. test |
|-------------|-----------|

Listing 11.1.8.4 Biochemical abnormalities at baseline. Grade  $\geq 2$ 

| Patient id | Parameter | Value | Units | Grade |
|------------|-----------|-------|-------|-------|

### 11.1.9 Coagulation Values at Baseline

Table 11.1.9.1 Coagulation abnormalities at baseline

| Tuoie 11:1:9:1 Congulation donormanties at ouseine | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | N | Gr | ade<br>1 | ••• | Gr | ade<br>4 | Al | 1* |
| | | N | % | | N | % | N | % |
| INR increased | | | | | | | | |
| PTT prolonged | | | | | | | | |

<sup>(\*)</sup>Any grade

Table 11.1.9.2 Coagulation values at baseline

| | N | Median | Min | Max |
|-----------|---|--------|-----|-----|
| INR | | | | |
| PT (sec) | | | | |
| PTT (sec) | | | | |

Listing 11.1.9.3 Coagulation tests not assessed at baseline

| Patient id. | Lab. test |
|-------------|-----------|

Listing 11.1.9.4 Coagulation abnormalities at baseline. Grade  $\geq 2$ 

| Patient id | Parameter | Value | Units | Grade |
|------------|-----------|-------|-------|-------|

# 11.1.10 Signs and Symptoms at Baseline

Table 11.1.10.1 Patients with signs and symptoms at baseline

| 5 , 1 | N | % |
|------------------------------------|---|---|
| No. signs and symptoms per patient | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥ 3 | | |
| Median (Range) | | |

Table 11.1.10.2 Patients with disease related signs and symptoms at baseline

| | N | % |
|-------------------------------------------------------|---|---|
| No. of disease related signs and symptoms per patient | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥ 3 | | |
| Median (Range) | | |

Table 11.1.10.3 Signs and symptoms at baseline

| SOC | Preferred Term | N | Gr | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|---|
| | | N | N | % | <br>N | % | N | % |
| Gastrointestinal disorders | Constipation | | | | | | | |
| | Diarrhea NOS | | | | | | | |

<sup>(\*)</sup>Any grade

Listing 11.1.10.4 Signs and Symptoms at baseline

| D-414-11 | Ci and for annual to an | C 1. * | 0 | D .1.41 |
|-------------|-------------------------|--------|------------|--------------|
| Patient id. | Sign/symptom | Grade* | Onset date | Relationship |
| l | | | | |

<sup>(\*)</sup>Those events with grade ≥ 2 or with relationship='Prior study disease treatment' will be highlighted.

# 11.1.11 Concomitant Therapy and Procedures at Baseline

Concomitant medication at baseline according to the ATC classification.

Table 11.1.11.1 Concomitant medication at baseline (ATC1/ATC2/ATC4/PN)

| Concomitant medication at baseline | N | % |
|------------------------------------|---|---|
| Alimentary tract and metabolism | | |
| Antacids | | |
| Magnesium compounds | | |
| Magnesium adipate | | |
| Blood and blood forming organs | | |
| Antithrombotic agents | | |
| Vitamin K antagonists | | |
| Acenocoumarol | | |

Table 11.1.11.2 Summary of concomitant medication at baseline

| | N | % |
|------------------------------------------|---|---|
| No. of systems at BL (ATC1 level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥3 | | |
| Median (range) | | |
| No. of indications at BL (ATC2 level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥ 3 | | |
| Median (range) | | |
| No. of agent families at BL (ATC4 level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥3 | | |
| Median (range) | | |

| | N | % |
|--------------------------------|---|---|
| No. of agents at BL (PN level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥3 | | |
| Median (range) | | |

Listing 11.1.11.3 Concomitant therapy

| | Patient | Туре | Agent/Procedure | Route | Daily<br>dose | Units | Start<br>date | Reason | Indication | Details | Start date of study drug administration |
|---|---|---|---|---|---|---|---|---|---|---|---|
| ١ | | | | | | | | | | | |

If there is a relevant number of patients receiving the same concomitant medication, a table summarizing this information might be added.

# 11.1.12Baseline and demographic characteristic comparisons

Table 11.1.12.1 Baseline and demographic characteristic comparisons by cohorts

| | | N | Cohort A | Cohort A1 | Cohort B | p-value* |
|---|---|---|---|---|---|---|
| Age | Median (range) | X | X.X (XX-XX) | X.X (XX-XX) | X.X (XX-XX) | X.XXXX |
| PS (ECOG) | 0 | X | X ( XX.X %) | X ( XX.X %) | X ( XX.X %) | X.XXXX |
| | 1 | | X ( XX.X %) | X ( XX.X %) | X ( XX.X %) | |
| BSA | Median (range) | | | | | |
| BRCA mutation | 1 | | | | | |
| | 2 | | | | | |
| Receptor status | Triple negative | | | | | |
| | HR+/HER2 - | | | | | |
| | HER2 + | | | | | |
| Liver metastases | Yes | | | | | |
| | No | | | | | |
| CNS metastases | Yes | | | | | |
| | No | | | | | |
| Sites involvement | <3 sites | | | | | |
| | ≥ 3 sites | | | | | |
| Advanced lines | Median (range) | | | | | |
| Advanced CT lines | Median (range) | | | | | |
| Prior Platinum | Yes | | | | | |
| | No | | | | | |
| Prior Anthracyclines | Yes | | | | | |

| | | N | Cohort A | Cohort A1 | Cohort B | p-value* |
|----------------------|-----|---|----------|-----------|----------|----------|
| | No | | | | | |
| Prior Taxanes | Yes | | | | | |
| | No | | | | | |
| Prior Capecitabine | Yes | | | | | |
| | No | | | | | |
| Prior PARP Inhibitor | Yes | | | | | |
| | No | | | | | |

<sup>\*</sup>Fisher's exact test (categorical variables);Mann-Whitney-Wilcoxon (continuous variables)

Table 11.1.12.2 Baseline and demographic characteristic comparisons: Platinum Yes/No in Cohort A

| | | N | Prior platinum<br>Yes | Prior platinum<br>No | p-value* |
|---|---|---|---|---|---|
| Age | Median (range) | X | X.X (XX-XX) | X.X (XX-XX) | X.XXXX |
| PS (ECOG) | 0 | X | X ( XX.X %) | X ( XX.X %) | X.XXXX |
| | 1 | | X ( XX.X %) | X ( XX.X %) | |

<sup>\*</sup>Fisher's exact test (categorical variables);Mann-Whitney-Wilcoxon (continuous variables). For the complete list of covarites, see table 11.1.12.1

Table 11.1.12.3 Baseline and demographic characteristic comparisons: BRCA 1 vs 2 in Cohort A

| | | N | BRCA 1 | BRCA 2 | p-value* |
|-----------|----------------|---|-------------|-------------|----------|
| Age | Median (range) | X | X.X (XX-XX) | X.X (XX-XX) | X.XXXX |
| PS (ECOG) | 0 | X | X ( XX.X %) | X ( XX.X %) | X.XXXX |
| | 1 | | X ( XX.X %) | X ( XX.X %) | |

<sup>\*</sup>Fisher's exact test (categorical variables);Mann-Whitney-Wilcoxon (continuous variables). For the complete list of covarites, see table 11.1.12.1

Table 11.1.12.4 Baseline and demographic characteristic comparisons: Prior PARPi Yes/No in Cohorts A+A1

| | | | Prior PARPi | Prior PARPi | |
|-----------|----------------|---|-------------|-------------|----------|
| | | N | Yes | No | p-value* |
| Age | Median (range) | X | X.X (XX-XX) | X.X (XX-XX) | X.XXXX |
| PS (ECOG) | 0 | X | X ( XX.X %) | X ( XX.X %) | X.XXXX |
| | 1 | | X ( XX.X %) | X ( XX.X %) | |

\*Fisher's exact test (categorical variables); Mann-Whitney-Wilcoxon (continuous variables). For the complete list of covarites, see table 11.1.12.1

Table 11.1.12.5 Baseline and demographic characteristic comparisons: Initial dose 7 mg FD vs 3.5 mg/m<sup>2</sup> in Cohort A

| | | N | 7 mg FD | 3.5 mg/m <sup>2</sup> | p-value* |
|---|---|---|---|---|---|
| Age | Median (range) | X | X.X (XX-XX) | X.X (XX-XX) | X.XXXX |
| PS (ECOG) | 0 | X | X ( XX.X %) | X ( XX.X %) | X.XXXX |
| | 1 | | X ( XX.X %) | X ( XX.X %) | |

<sup>\*</sup>Fisher's exact test (categorical variables); Mann-Whitney-Wilcoxon (continuous variables). For the complete list of covarites, see table 11.1.12.1

Table 11.1.12.6 Baseline and demographic characteristic comparisons: Hormonal status triple negative vs Other

| triple negativ | • 15 5 11101 | | | | |
|---|---|---|---|---|---|
| | | N | Triple negative<br>Yes | Triple negative<br>No | p-value* |
| Age | Median (range) | X | X.X (XX-XX) | X.X (XX-XX) | X.XXXX |
| PS (ECOG) | 0 | X | X ( XX.X %) | X ( XX.X %) | X.XXXX |
| | 1 | | X ( XX.X %) | X ( XX.X %) | |

<sup>\*</sup>Fisher's exact test (categorical variables); Mann-Whitney-Wilcoxon (continuous variables). For the complete list of covarites, see table 11.1.12.1

Table 11.1.12.7 Baseline and demographic characteristic comparisons: Advanced chemotherapy lines

| | | N | 0-1 lines | >1 lines | p-value* |
|-----------|----------------|---|-------------|-------------|----------|
| Age | Median (range) | X | X.X (XX-XX) | X.X (XX-XX) | X.XXXX |
| PS (ECOG) | 0 | X | X ( XX.X %) | X ( XX.X %) | X.XXXX |
| | 1 | | X ( XX.X %) | X ( XX.X %) | |

<sup>\*</sup>Fisher's exact test (categorical variables); Mann-Whitney-Wilcoxon (continuous variables). For the complete list of covarites, see table 11.1.12.1

### 11.2 Measurements of Treatment Compliance

Compliance of individual patients with the treatment regimen under study will be measured and tabulated in section 12.1 and listed in appendix 16.2.5 (ICH listings).

### 11.3 Efficacy Analysis

Efficacy analysis will be carried out on the "All Evaluable Patients" population.

Subgroup analysis will be performed in Cohort A according to prior treatment with platinum, BRCA status (BRCA1 vs. BRCA2), hormonal status (Triple negative vs. HR+), number of advanced chemotherapy lines , prior PARPi (Yes vs. No) and starting dose (7 mg FD vs. 3.5 mg/m²).

Subgroup analysis will be performed in Cohorts A+A1 according to prior PARPi (Yes vs. No).

The tables included in each subgroup analysis are the following:

Table 11.3.1.1 Response rate

Table 11.3.1.2 Overall response rate

Table 11.3.2.1 Duration of response

Table 11.3.2.2 Progression-free survival (PFS)

Table 11.3.2.3 Overall survival (OS)

The tables will be annotated by adding a letter as suffix:

- BRCA status: a

- Prior platinum: b

- Hormonal status: c

- Advanced chemotherapy lines: d

- Starting dose: e

- Prior PARPi (Cohort A): f

- Prior PARPi (Cohorts A+A1): g

If any other disease characteristic is sufficiently represented and clinically relevant, subgroup analysis may be performed, and their corresponding tables will also be annotated by adding a letter to the table's name.

#### 11.3.1 Primary Analysis

Table 11.3.1.1 Response rate

| Tuote 11.5.1.1 Response tute | | |
|------------------------------|---|---|
| Response | N | % |
| Complete response (CR) | | |
| Partial response (PR) | | |
| Stable disease (SD) | | |
| Progressive disease (PD) | | |
| Inevaluable for efficacy* | | |

<sup>(\*)</sup> Treatment failures

Table 11.3.1.2 Overall response rate

| | Proportion | Lower 95% limit | Upper 95% limit |
|----------------|------------|-----------------|-----------------|
| Response rate* | | | |

(\*) CR + PR

Binomial exact estimator and 95% CI

# 11.3.2 Secondary Analysis

Table 11.3.2.1 Duration of response (DR)

| | DR |
|-----------------|----|
| N | |
| Events | |
| Censored | |
| Median DR | |
| DR at 6 months | |
| DR at 12 months | |

Kaplan-Meier plot will be also shown (Figure 11.3.2.1)

Table 11.3.2.2 Progression-free survival (PFS)

| | PFS |
|------------------|-----|
| N | |
| Events | |
| Censored | |
| Median PFS | |
| PFS at 3 months | |
| PFS at 6 months | |
| PFS at 12 months | |

Kaplan-Meier plot will be also shown (Figure 11.3.2.2)

### Table 11.3.2.3 Overall survival (OS)

| | OS |
|-----------------|----|
| N | |
| Events | |
| Censored | |
| Median OS | |
| OS at 12 months | |
| OS at 18 months | |

Kaplan-Meier plot will be also shown (Figure 11.3.2.3)

### Table 11.3.2.4 Clinical benefit rate

| | Proportion | Lower 95% limit | Upper 95% limit |
|------------------------|------------|-----------------|-----------------|
| Clinical benefit rate* | | | |

(\*) CR + PR + SD > 3 months

Binomial exact estimator and 95% CI

Listing 11.3.2.5 Characteristics of patients with clinical benefit\*.

| | • | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient | | PS / | BRCA | Histology | Histology | Hormonal<br>Status | ıs | No.<br>of<br>prior | No. of advanced CT lines | Prior<br>Platinum<br>(Y/N) | Best<br>response<br>Prior | Prior last therapy | |
| | Age | status | Type | Grade | | Sites | lines | | | platinum | Agents | Best<br>response | PFS<br>(months |
| | ! | | | | | | | | | | | | |

(\*) CR + PR + SD > 3 months
| Patient | Initial dose | Cycles received | Best response | PFS (months) | OS<br>(months) | DR (months) |
|---|---|---|---|---|---|---|

<sup>(\*)</sup> CR + PR + SD > 3 months

Table 11.3.2.6 Median follow-up\*

| | T-F | |
|-----------|--------|--------|
| Follow-up | Median | 95% CI |
| PFS | | |
| OS | | |

<sup>\*</sup>Calculated using the Kaplan-Meier method reversing the censoring values.

Figure 11.3.2.7 "Waterfall plot" ΔSum of lesions from BL



Figure 11.3.2.8 "Swimmer plot" PFS in Cohort A



Figure 11.3.2.9 "Swimmer plot" PFS in Cohort A1



Figure 11.3.2.10 "Swimmer plot" PFS in Cohort B



## 11.3.3 Exploratory Univariate and Multivariate Analyses

Table 11.3.3.1 Univariate analysis of response rate

| | | | | | 1 | | | |
|---|---|---|---|---|---|---|---|---|
| Variable<br>label | Variable values | DF | Estimate | Standard<br>error | Wald chi-<br>square | Pr > ChiSq | ( )dde ratio | 95% Odds Ratio<br>confidence<br>limits |

(See list of covariates in section 6.2.2).

Table 11.3.3.2 Multivariate analysis of response rate

| | Analysis of Maximum Likelihood Estimates | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable<br>label | Variable values | DF | Estimate | Standard<br>error | Wald chi-<br>square | Pr > ChiSq | Odds ratio estimate | 95% Odds Ratio<br>confidence<br>limits |

(See list of covariates in section 6.2.2. Only those covariates with a p-value < 0.10 in univariate analysis and with a 90% of valid observations will be included).

Table 11.3.3.3 Univariate analysis of PFS

| Variable label | Variable values | DF | Parameter estimate | Standard<br>error | Chi-square | Pr > ChiSq | Hazard<br>ratio | 95% Hazard ratio confidence limits |
|---|---|---|---|---|---|---|---|---|

(See list of covariates in section 6.2.2).

Table 11.3.3.4 Multivariate analysis of PFS

| | Analysis of Maximum Likelihood Estimates | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable label | Variable values | DF | Parameter estimate | Standard<br>error | Chi-square | Pr > ChiSq | Hazard<br>ratio | 95% Hazard ratio confidence limits |

(See list of covariates in section 6.2.2. Only those covariates with a p-value < 0.10 in univariate analysis and with a 90% of valid observations will be included).

Table 11.3.3.5 Univariate analysis of OS

| Variable label | Variable values | DF | Parameter estimate | Standard error | Chi-square | Pr > ChiSq | Hazard<br>ratio | 95% Hazard ratio confidence limits |
|---|---|---|---|---|---|---|---|---|

(See list of covariates in section 6.2.2).

Table 11.3.3.6 Multivariate analysis of OS

| | Analysis of Maximum Likelihood Estimates | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable label | Variable values | DF | Parameter estimate | Standard<br>error | Chi-square | Pr > ChiSq | Hazard<br>ratio | 95% Hazard ratio confidence limits |

(See list of covariates in section 6.2.2. Only those covariates with a p-value < 0.10 in univariate analysis and with a 90% of valid observations will be included).

# 12 Safety Analysis

Safety analysis will be carried out on the "All Treated Patients" population.

#### 12.1 Extent of Exposure

Subgroup analysis will be performed according to starting dose (7 mg FD vs. 3.5 mg/m<sup>2</sup>). The tables will be annotated by adding a letter as suffix.

The tables included in the subgroup analysis are the following:

Table 12.1.1.1 Number of cycles administered and dose intensity

Table 12.1.2.1.3 Number of patients and cycles with dosing delay according to relationship

Table 12.1.3.3 Number of patient and cycles with dose reduction according to relationship

## 12.1.1 Treatment Administration

Table 12.1.1.1 Number of cycles administered and dose intensity

| No. of cycles administered per patient | N | % |
|----------------------------------------|---|---|
| 1 | | |
| 2 | | |
| 3 | | |
| Median (range) | | • |
| Time on treatment* (weeks) | | |
| Median | | |
| Range | | |
| PM01183 cumulative dose (mg) | | |
| Median | | |
| Range | | |
| PM01183 dose intensity (mg/wk) | | |
| Median | | |
| Range | | |
| PM01183 relative dose intensity (%) | | |
| Median | | |
| Range | | |

<sup>(\*)</sup>Time on treatment: defined as last infusion date plus 30 days, or date of death or subsequent therapy (whichever comes first) minus first infusion date.

#### 12.1.2 Cycle Delays

## 12.1.2.1 Number of Patients and Cycles with Dosing Delay, Any Relationship

Listing 12.1.2.1.1 Delays

| ] | Patient id. | Delayed<br>cycle | Delayed<br>cycle start<br>date | Previous cycle | Previous cycle start date | Dose Delay calculated. (days) | Reason for dose delay | Dose Delay<br>Spec. |
|---|---|---|---|---|---|---|---|---|

Table 12.1.2.1.2 Number of patients and cycles with dosing delay, any relationship

| | N | % |
|------------------------------------------------------|---|---|
| No. of patients treated | | |
| No. of patients susceptible to have any dose delayed | | |
| No. of patients with any dose delayed | | |
| No. of cycles administered | | |
| No. of cycles susceptible to be delayed* | | |
| No. of cycles with dosing delay** | | |
| No. of patients with | | |
| No cycles delayed | ļ | |
| 1 cycle delayed | ļ | |
| 2 cycles delayed | | |
| ≥ 3 cycles delayed | ļ | |

<sup>(\*)</sup> All cycles excluding first cycle. (\*\*) Denominator= Number of cycles susceptible to be delayed

Table 12.1.2.1.3 Number of patients and cycles with dosing delay according to the relationship

| _ | Treatme | ent-related** | Non-treatment-related | |
|---|---|---|---|---|
| | N | % | N | % |
| No. of patients with 1 cycle delayed 2 cycles delayed ≥ 3 cycles delayed | | | | |
| No. of cycles with dosing delay* | | | | |

<sup>(\*)</sup> Denominator= Number of cycles susceptible to be delayed. (\*\*)Hematological reason, non-hematological reason or both

Table 12.1.2.1.4 Number of patients and cycles with dosing delay according to the relationship

| Reasons f | or delays | N | % |
|-----------|-------------------------------------|---|------|
| Cycles | No. of cycles with dosing delays* | | • |
| | Treatment-related | X | XX.X |
| | Hematological | | |
| | Non-hematological | | |
| | Both | | |
| | Non-treatment-related | | |
| Patients | No. of patients with dosing delays* | | |
| | Treatment-related | X | XX.X |
| | Hematological | | |
| | Non-hematological | | |
| | Both | | |
| | Non-treatment-related | | |

<sup>(\*)</sup> Denominator= Number of patient/cycles susceptible to have a delay.

Table 12.1.2.1.5 Length of dosing delay.

| | Treatment-related** | | Non-treatr | Total | | |
|---|---|---|---|---|---|---|
| Length of delay Median (range) | | | | | | |
| Length of delay* | N | % | N | % | N | % |
| <= 7 days | | | | | | |
| >7 days and <=14 days | | | | | | |
| > 14 days | | | | | | |

<sup>(\*)</sup> Denominator= Number of cycles susceptible to be delayed. (\*\*)Hematological reason, Non-hematological reason or both

## 12.1.2.2 Number of Delays According to Cycle Number

Table 12.1.2.2.1 Number and reasons of delays according to cycle number

| Tweeto 12.11,2.211 Tyunne of which found in the control of weiting the open manne of | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | No. of No. of | | | | ment- | Treatment-related | | | | | | Non- | | |
| | | | del | delays related* | | Hematological reason Non-hematological reason | | Both | | treatment-<br>related* | | | | |
| | N | % | N | % | N | % | N | % | N | % | N | % | N | % |
| Cycle 2 | | | | | | | | | | | | | | |
| Cycle 6 | | | | | | | | | | | | | | |

<sup>(\*)</sup> Denominator= Number of cycles susceptible to be delayed.

Table 12.1.2.2.2 Dose reduction in cycles delayed

| | | Reduction | | |
|---------|---|-----------|---|----|
| | , | Yes | ] | No |
| | N | % | N | % |
| Cycle 2 | | | | |
| Cycle 6 | | | | |
| ••• | | | | |
| Total | | | | |

The distribution of delays according to the cycle administered will be studied by means of counts and percentages. The reasons for cycle delay will be detailed, specifying how many were due to treatment or not.

Listing 12.1.2.2.3 Cycle delays due to AEs

| Patient id. | CVCLE | Preferred<br>term code | Adverse<br>event<br>reported<br>(verbatim) | Relationship | Onset<br>date | Resolved<br>date | No. of days with delay | Action taken | Significant consequences |
|---|---|---|---|---|---|---|---|---|---|

AEs with action = 'Dose delayed' or 'Reduced and delayed'.

#### 12.1.3 Dose Reductions

All dose reductions should be considered and described, specifying the reason for reduction (hematological toxicity, non-hematological toxicity or other causes).

Listing 12.1.3.1 Dose reductions

| Patient id. | Cycle | Day | Cycle start date | Previous dose | Reduced dose | Reason for dose reduction | Dose reduction Spec. |
|---|---|---|---|---|---|---|---|

Table 12.1.3.2 Number of patients and cycles with dose reduction, any relationship

| | N | % |
|---------------------------------------------------------------|---|------|
| No. of patients treated | X | XX.X |
| No. of patients susceptible to have a dose reduced | | |
| No. of patients with any dose reduced | | |
| No. of patients with: | | |
| No PM01183 reduction | | |
| 1 cycle with PM01183 dose reduced | | |
| 2 cycles with PM01183 dose reduced | | |
| No. of cycles administered | | |
| No. of cycles susceptible to have any dose reduced* | | |
| No. of cycles with PM01183 dose reduced ** | | |
| No. of cycles with PM01183 dose reduced (Treatment-related)** | | |

<sup>(\*)</sup> All cycles excluding first cycle. (\*\*) Denominator= Number of cycles susceptible to have a dose reduction

Table 12.1.3.3 Number of patients and cycles with dose reduction according to the relationship

| Reasons for r | eductions | N | % |
|---------------|---------------------------------------|---|------|
| Cycles | No. of cycles with dose reductions* | | |
| | Treatment-related | X | XX.X |
| | Hematological | | |
| | Non-hematological | | |
| | Both | | |
| | Non-treatment-related | | |
| Patients | No. of patients with dose reductions* | | |
| | Treatment-related | X | XX.X |
| | Hematological | | |
| | Non-hematological | | |
| | Both | | |
| | Non-treatment-related | | |

<sup>(\*)</sup> Denominator= Number of patient/cycles susceptible to have a dose reduction.

Table 12.1.3.4 Number and reasons of reductions according to cycle number

| | No. of cycles patients with | | with related* | | Treatment-related | | | | | | Non-<br>treatment- | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | ieu · | Hematological reason | | Non-<br>hematological<br>reason | | Both | | related* | | |
| | N | % | N | % | N | % | N | % | N | % | N | % | N | % |
| Cycle 1<br>Cycle 2 | | | | | | | | | | | | | | |
| Cycle 6 | | | | | | | | | | | | | | |

<sup>(\*)</sup> Denominator= Number of cycles susceptible to be reduced.

Listing 12.1.3.5 Dose reductions due to AEs

| Patient id. | Total<br>no. of<br>cycles | Cycle | Preferred term code | Adverse<br>event<br>reported<br>(verbatim) | Relationship | Onset<br>date | Resolved date | Action taken | Significant consequences |
|---|---|---|---|---|---|---|---|---|---|

AEs with action = 'Dose reduced/adjusted' or 'Reduced and delayed'.

#### 12.1.4 Infusions Temporarily Interrupted

A listing of the patients who had infusions temporarily interrupted with the corresponding reasons will be provided.

Listing 12.1.4.1 Interrupted infusion listing.

| Patient id. | Cycle | Reason |
|-------------|-------|--------|

## 12.1.5 Prophylactic Medication Administration

A listing of the patients who have not received corticosterioids, 5-HT antagonists, prokinetics and other antiemetics or equivalents with the corresponding reasons will be reported.

Listing 12.1.5.1 Patients and cycles with prophylactic medication not taken per protocol

| Patient id. | Cycle | Prophylactic medication not | Reason |
|-------------|-------|-----------------------------|--------|
| | | taken* | |
| | | No | |

<sup>(\*)</sup> Corticosterioids, 5-HT antagonists, prokinetics and other antiemetics.

#### 12.2 Adverse Events

#### 12.2.1 Adverse Events

As far as all the toxicities are concerned, the NCI-CTC grade will be used wherever an NCI-CTC grading exists. Otherwise, the severity will be noted. As a convention, the term «Grade» will always be used. Toxicities will be described according to the worst NCI-CTC grade or, for toxicities which do not form the subject of NCI-CTC classification, according to the worst severity.

Adverse events will be described in this section; treatment-related events (stated as related to the study drug or of unknown relationship) will be tabulated.

Type of toxicity and worst grade or severity by cycle and by patient will be summarized according to the Preferred Term coded with MedDRA. Tables will be organized per category of events using System Organ Class of MedDRA.

Subgroup analysis will be performed according to starting dose (7 mg FD vs. 3.5 mg/m2) and Cohort.

The groups will include:

- Patient treated at 7 mg FD Cohort B
- Patient treated at 7 mg FD Cohort A
- Patient treated at 7 mg FD any Cohort
- Patient treated at 3.5 mg/m<sup>2</sup> Cohort A
- Patient treated at 3.5 mg/m<sup>2</sup> Cohort A1
- Patient treated at 3.5 mg/m<sup>2</sup> any Cohort

The tables will be annotated by adding a letter as suffix.

The tables included in the subgroup analysis are the following:

Table 12.2.2.2 Treatment related AEs. Worst grade by patient

Table 12.2.2.3 Treatment related AEs. Worst grade by cycle

Table 12.2.2.4 Adverse events regardless of relationship. Worst grade by patient

Table 12.2.2.5 Adverse events regardless of relationship. Worst grade by cycle

If clinically relevant the outputs could be split by initial dose or any other characteristic.

# 12.2.2 Display of Adverse Events

Table 12.2.2.1 Summary of AEs.

| Category | N | % |
|------------------------------------------------------------|---|---|
| Patients with at least one AE regardless relationship | | |
| Any treatment-related AE | | |
| Any grade 3/4 AE | | |
| Any grade 3/4 treatment-related AE | | |
| Any SAE in DB | | |
| Any treatment-related SAE | | |
| Any grade 3/4 SAE | | |
| Any grade 3/4 treatment-related SAE | | |
| AEs leading to death | | |
| AEs treatment-related leading to death | | |
| AEs leading to dose delay | | |
| AEs leading to dose reduction | | |
| AEs leading to treatment discontinuation | | |
| AEs treatment-related leading to treatment discontinuation | | |

Table 12 2 2 2 Treatment-related AEs Worst grade by natient

| 14010 12.2.2.2 1104 | timent related ribb. We orbit | 5raac oj | Patron | · | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | Gr | Grade<br>1 | | Grade<br>1 | | Gr | ade<br>4 | A | 11* |
| | | N | % | | N | % | N | % | | |
| Blood and lymphatic system disorders | Anemia NOS | | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.2.2.3 Treatment-related AEs. Worst grade by cycle

| SOC | SOC Preferred Term Grade 1 | | Grade<br>1 | Grade<br>1 | | Grad | | A | 11* |
|---|---|---|---|---|---|---|---|---|---|
| | | N | % | N | % | N | % | | |
| Blood and lymphatic system disorders | Anemia NOS | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | | |

<sup>\*</sup> Any grade

Table 12.2.2.4 Adverse Events regardless of relationship. Worst grade by patient

| SOC | Preferred Term | Grade<br>1 | | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|
| | | N | % | <br>N | % | N | % |
| Blood and lymphatic system disorders | Anemia NOS | | | | | | |
| System disorders | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.2.2.5 Adverse Events regardless of relationship. Worst grade by cycle

| SOC | Preferred Term | Grade<br>1 | | Grade 4 | | ade<br>4 | All* | |
|---|---|---|---|---|---|---|---|---|
| | | N | % | | N | % | N | % |
| Blood and lymphatic system disorders | Anemia NOS | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | |

<sup>(\*)</sup> Any grade

Listing 12.2.2.6 Treatment-related grade 3-4 AEs. Worst grade per patient

| Patient id. | SOC Name | Preferred term | Grade |
|-------------|----------|----------------|-------|

Listing 12.2.2.7 Treatment-related grade 3-4 AEs. Worst grade by cycle

| Patient id. | Cycle | SOC Name | Preferred term | Grade |
|-------------|-------|----------|----------------|-------|

# Listing 12.2.2.8 Adverse Events grade 3-4 regardless of relationship. Worst grade per patient

| Patient id. | SOC Name | Preferred term | Grade |
|-------------|----------|----------------|-------|

Listing 12.2.2.9 Adverse Events grade 3-4 regardless of relationship. Worst grade by cycle

| _ | 0 | | | | |
|---|-------------|-------|----------|----------------|-------|
| | Patient id. | Cycle | SOC Name | Preferred term | Grade |
| F | | | | | |

Table 12.2.2.10 Treatment-related SAEs. Worst grade by patient

| SOC | Preferred Term | Grade<br>1 | | Grade<br>1 | | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|---|---|
| | | N | % | <br>N | % | N | % | | |
| Blood and lymphatic | Anemia NOS | | | | | | | | |
| system disorders | | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.2.2.11 Treatment-related SAEs. Worst grade by cycle

| SOC | Preferred Term | Grade<br>1 | | Grade<br>1 | | Grade<br>1 | | Grade<br>1 | Grade<br>1 | Grade<br>1 | Grade<br>1 | Grade<br>1 | Grade<br>1 | Grade<br>1 | Grade<br>1 | Grade<br>1 | Grade<br>1 | Grade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | N | % | <br>N | % | N | % | | | | | | | | | | | | | | | |
| Blood and lymphatic | Anemia NOS | | | | | | | | | | | | | | | | | | | | | |
| system disorders | | | | | | | | | | | | | | | | | | | | | | |

| Cardiac disorders | Arrhythmia NOS |
|-------------------|----------------|

<sup>\*</sup> Any grade

Table 12.2.2.12 SAEs regardless of relationship. Worst grade by patient

| SOC | Preferred Term | Grade<br>1 | | <br>Grade<br>4 | | All* | |
|---|---|---|---|---|---|---|---|
| | | N | % | <br>N | % | N | % |
| Blood and lymphatic | Anemia NOS | | | | | | |
| system disorders | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.2.2.13 SAEs regardless of relationship. Worst grade by cycle

| SOC | Preferred Term | | Grade<br>1 | Grade 4 | | All* | |
|---|---|---|---|---|---|---|---|
| | | N | % | N | % | N | % |
| Blood and lymphatic | Anemia NOS | | | | | | |
| system disorders | ••• | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | |

<sup>(\*)</sup> Any grade

At the time of the analysis, if appropriate, grouping of similar or clinically related items will be made.

# 12.2.3 Evolution of signs and symptoms during the treatment

Worst grade signs and symptoms present during treatment and at baseline regardless of relationship will be shown.

Table 12.2.3.1 Shift of signs and symptoms during the treatment

| | | Worst grade per patient during treatment | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| MedDRA PT | Baseline grade | Grade<br>1 | | Grade Grade 1 2 | | Grade 3 | | Grade<br>4 | |
| | | N | % | N | % | N | % | N | % |
| Constipation | 1 | | | | | | | | |
| | 2 | | | | | | | | |
| | ••• | | | | | | | | |
| Diarrhea | 1 | | | | | | | | |
| | 2 | | | | | | | | |
| | ••• | | | | | | | | |

#### 12.3 Serious Adverse Events and Deaths.

## 12.3.1 Serious Adverse Events

Listing 12.3.1.1 SAEs

| Patient id. | Preferred term code | Adverse event reported (verbatim) | Grade | Relationship | Onset<br>date | Resolved<br>date | Action | Serious criteria |
|---|---|---|---|---|---|---|---|---|

The Pharmacovigilance Department will provide the narratives of the SAEs from the Pharmacovigilance Database (DB).

#### 12.3.2 Deaths

#### Table 12.3.2.1 Cause of death

| Reason* | N | % |
|----------------------------------|---|---|
| Malignant disease | | |
| Study drug related adverse event | | |
| Non-study drug related AE | | |
| Other | | |
| Total | | |

<sup>(\*)</sup> Denominator=Number of patients who died

#### Listing 12.3.2.2 Deaths

| Patie<br>id. | Death date | Cause | Comments | Autopsy | Number of cycles administered | Last infusion date | Time on treatment* | Time from<br>Last dose** |
|---|---|---|---|---|---|---|---|---|

<sup>(\*)</sup>Time on treatment: defined as last infusion date plus 30 days, or date of death or subsequent therapy (whichever comes first) minus first infusion date. (\*\*)Time from last dose defined as death date minus last infusion date.

### Listing 12.3.2.3 AEs with outcome death

| Patient id. | Cycle | Preferred term code | Adverse event reported (verbatim) | Grade | Relationship | Onset<br>date | Date of death | Action |
|---|---|---|---|---|---|---|---|---|

#### 12.4 Clinical Laboratory Evaluation

Subgroup analysis will be performed according to starting dose (7 mg FD vs. 3.5 mg/m<sup>2</sup>) and Cohort.

The groups will include:

- Patient treated at 7 mg FD Cohort B
- Patient treated at 7 mg FD Cohort A
- Patient treated at 7 mg FD any Cohort
- Patient treated at 3.5 mg/m<sup>2</sup> Cohort A
- Patient treated at 3.5 mg/m<sup>2</sup> Cohort A1
- Patient treated at 3.5 mg/m<sup>2</sup> any Cohort

The tables will be annotated by adding a letter as suffix.

The tables included in the subgroup analysis are the following:

- Table 12.4.1.1 Hematological abnormalities during treatment, worst grade per patient
- Table 12.4.1.2 Hematological abnormalities during treatment, worst grade per cycle
- Table 12.4.2.1 Biochemical abnormalities during treatment, worst grade per patient
- Table 12.4.2.2 Biochemical abnormalities during treatment, worst grade per cycle
- Table 12.4.3.1 Coagulation abnormalities during treatment, worst grade per patient
- Table 12.4.3.2 Coagulation abnormalities during treatment, worst grade per cycle

## 12.4.1 Hematological Abnormalities

Hematological toxicities classified according to the NCI-CTC will be calculated for all cycles. The worst grade reached by each patient during treatment will be also calculated.

If serious toxicities happen, special follow-up, with descriptives and graphs (boxplots, line plots), will be made to find out the pattern of thrombocytopenia and neutropenia within and between the different cycles.

Table 12.4.1.1 Hematological abnormalities during treatment, worst grade per patient

| | Grade | | Grade<br>4 | | All* | | | |
|------------------|-------|---|------------|-----|------|---|---|---|
| | | N | % | ••• | N | % | N | % |
| Leukopenia | | | | | | | | |
| Anemia | | | | | | | | |
| Thrombocytopenia | | | | | | | | |
| Neutropenia | | | | | | | | |
| Lymphopenia | | | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.4.1.2 Hematological abnormalities during treatment, worst grade per cycle

| | N | Gr | ade<br>1 | | Gra | ade<br>1 | Al | 1* |
|------------------|---|----|----------|-----|-----|----------|----|----|
| | | N | % | ••• | N | % | N | % |
| Leukopenia | | | | | | | | |
| Anemia | | | | | | | | |
| Thrombocytopenia | | | | | | | | |
| Neutropenia | | | | | | | | |
| Lymphopenia | | | | | | | | |

<sup>(\*)</sup> Any grade

Listing 12.4.1.3 Grade 3-4 hematological abnormalities during treatment. Worst grade per patient

| Patient id. | Cycle | Test | Grade |
|-------------|-------|------|-------|

Listing 12.4.1.4 Grade 3-4 hematological abnormalities during treatment. Worst grade per cycle

| Patient id. | Cycle | Test | Grade |
|-------------|-------|------|-------|

Listing 12.4.1.5 Hematological tests not assessed by patient and cycle

| Patient id. | Cycle | Lab. test |
|-------------|-------|-----------|

#### 12.4.2 Biochemical Abnormalities

Grades of liver toxicity and intercycle pattern of creatinine, CPK, bilirubin, transaminases increase and alkaline phosphatase increase during a cycle will be calculated, as it is explained in the section 7.2 for biochemical toxicities.

Table 12 4 2 1 Biochemical abnormalities during treatment, worst grade per patient

| <br> | 2 0,000 | <br>8 p p | |
|------|---------|-----------|------|
| N | Grade | <br>Grade | All* |

| | | 1 | | 4 | | | |
|---------------------------|---|---|-------|---|---|---|---|
| | N | % | • • • | N | % | N | % |
| AST increased | | | | | | | |
| ALT increased | | | | | | | |
| Total bilirubin increased | | | | | | | |
| AP increased | | | | | | | |
| Hyperglycemia | | | | | | | |
| Hypoglycemia | | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.4.2.2 Biochemical abnormalities during treatment, worst grade per cycle

| | N | Grade<br>1 | | <br>Grade 4 | | All* | |
|---------------------------|---|------------|---|-------------|---|------|---|
| | | N | % | <br>N | % | N | % |
| AST increased | | | | | | | |
| ALT increased | | | | | | | |
| Total bilirubin increased | | | | | | | |
| AP increased | | | | | | | |
| Hyperglycemia | | | | | | | |
| Hypoglycemia | | | | | | | |

<sup>(\*)</sup> Any grade

Listing 12.4.2.3 Grade 3-4 biochemical abnormalities during treatment. Worst grade per patient

| Patient id. | Cycle | Test | Grade |
|-------------|-------|------|-------|

Listing 12.4.2.4 Grade 3-4 biochemical abnormalities during treatment. Worst grade per cycle

| Patient id. | Cycle | Test | Grade |
|-------------|-------|------|-------|

Listing 12.4.2.5 Biochemical tests not assessed by patient and cycle

| г | <u> </u> | J I | <u> </u> |
|---|-------------|-------|-----------|
| | Patient id. | Cycle | Lab. test |
| ſ | | | |

# 12.4.3 Coagulation Abnormalities

Table 12.4.3.1 Coagulation abnormalities during treatment, worst grade per patient

| | N | Grad<br>N 1 | | Grade | | ade<br>3 | All* | |
|----------------|---|-------------|---|-------|---|----------|------|---|
| | | N | % | | N | % | N | % |
| INR increased | | | | | | | | |
| APTT prolonged | | | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.4.3.2 Coagulation abnormalities during treatment, worst grade per cycle

| | N | Grade<br>1 | | <br>Grade<br>3 | | All* | |
|----------------|---|------------|---|----------------|---|------|---|
| | | N | % | <br>N | % | N | % |
| INR increased | | | | | | | |
| APTT prolonged | | | | | | | |

<sup>(\*)</sup> Any grade

Listing 12.4.3.3 Grade 3 coagulation abnormalities during treatment. Worst grade per patient

| r | | | |
|-------------|-------|------|-------|
| Patient id. | Cycle | Test | Grade |

## Listing 12.4.3.4 Grade 3 coagulation abnormalities during treatment. Worst grade per cycle

| 21011116 12:::011 | | | . Herst Bruss per ejere |
|-------------------|-------|------|-------------------------|
| Patient id. | Cycle | Test | Grade |

Listing 12.4.3.5 Coagulation tests not assessed by patient and cycle

| | <i>J</i> 1 | J |
|-------------|------------|-----------|
| Patient id. | Cycle | Lab. test |

## 12.4.4 Laboratory Values Over Time

In this section, grades 3-4 hematological and liver enzyme abnormalities will be displayed according to the cycle in which they occurred.

Table 12.4.4.1 Evolution of hematological abnormalities from baseline, worst case per patient.

| | | Baseline grade* | | V | orst gra | ade per p | atient | | т | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 0 | | 1 | | | 1 | otai |
| | | | N | % | N | % | N | % | N | % |
| | Neutropenia | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| | Thrombocytopenia Grade 0 | | | | | | | | | |
| ine | | Grade 0 | | | | | | | | |
| Baseline | | Grade 1 | | | | | | | | |
| Ba | | | | | | | | | | |
| | | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |

<sup>\*</sup>Defined as the last value recorded before or on the date of first infusion.

Table 12.4.4.2 Evolution of hematological abnormalities from baseline, worst case in the

first cycle per patient.

| | | | V | Vorst gra | de in th | e first cy | cle per p | atient | т | otal |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Baseline grade* | | 0 | | 1 | | | Total | |
| | | | N | % | N | % | N | % | N | % |
| | Neutropenia Grade 0 | | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| ine | Thrombocytopenia | Grade 0 | | | | | | | | |
| Baseline | | Grade 1 | | | | | | | | |
| Ba | | | | | | | | | | |
| | •••• | Grade 0<br>Grade 1 | | | | | | | | |

<sup>\*</sup>Defined as the last value recorded before or on the date of first infusion.

Table 12.4.4.3 Evolution of hematological abnormalities from baseline, worst case in the last cycle per patient.

| | | | W | orst gra | de in th | e last cyc | ele per pa | tient | т. | n+n1 |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Baseline grade* | | 0 | | 1 | | | Total | |
| | | | N | % | N | % | N | % | N | % |
| | Neutropenia | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| ine | Thrombocytopenia | Grade 0 | | | | | | | | |
| Baseline | | Grade 1 | | | | | | | | |
| Ba | | | | | | | | | | |
| | | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |

<sup>\*</sup>Defined as the last value recorded before or on the date of first infusion.

Table 12.4.4.4 Evolution of biochemical abnormalities from baseline, worst case per

patient.

| | | | | V | , | Γotal | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Baseline grade* | | 0 | | 1 | | | - | otai |
| | | | N | % | N | % | N | % | N | % |
| | AST increase | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| ine | ALT increase | Grade 0 | | | | | | | | |
| Baseline | | Grade 1 | | | | | | | | |
| Ba | | | | | | | | | | |
| | | Grade 0 | | | | | | | | |
| | Grade 1 | | | | | | | | | |

<sup>\*</sup>Defined as the last value recorded before or on the date of first infusion.

Table 12.4.4.5 Evolution of biochemical abnormalities from baseline, worst case in the first

cycle per patient.

| | | | | Worst g | rade in t | first cycl | e per pa | tient | - | Cotol |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Baseline grade* | | 0 | | 1 | | | Total | |
| | | N | N | % | N | % | N | % | N | % |
| | AST increase Grade 0 | | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| ine | ALT increase | Grade 0 | | | | | | | | |
| Baseline | | Grade 1 | | | | | | | | |
| $\mathbf{Ba}$ | | | | | | | | | | |
| | | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |

<sup>\*</sup>Defined as the last value recorded before or on the date of first infusion.

Table 12.4.4.6 Evolution of biochemical abnormalities from baseline, worst case in last

cycle per patient.

| | • | | | Worst g | rade in | last cycle | e per pat | ient | т | oto1 |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Baseline grade* N | | 0 | | 1 | | | Total | |
| | | | N | % | N | % | N | % | N | % |
| | AST increase | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| ine | ALT increase | Grade 0 | | | | | | | | |
| Baseline | | Grade 1 | | | | | | | | |
| Ва | | | | | | | | | | |
| | | Grade 0<br>Grade 1 | | | | | | | | |

<sup>\*</sup>Defined as the last value recorded before or on the date of first infusion.

Table 12.4.4.7 Grade 3-4 laboratory abnormalities in the first cycle and in all other cycles

| Laboratory | Cycle 1 | | | Cycle>1 | | |
|---|---|---|---|---|---|---|
| Laboratory abnormalities | No. of cycles evaluated | No. of cycles grade 3-4 | % | No. of cycles evaluated | No. of cycles grade 3-4 | % |
| Thrombocytopenia | | | | | | |
| AP | | | | | | |
| Total bilirubin | | | | | | |
| AST | | | | | | |
| ALT | | | | | | |
| СРК | | | | | | |

Listing 12.4.4.8 Summary of grade 4 neutropenia and G-CSF administration

| Patient | Total number of cycles | Cycle numbers with grade 4 | Cycle numbers with G-CSF | Cycle numbers with |
|---|---|---|---|---|
| 1 attent | received | neutropenia | administration | dose reduction |

Listing 12.4.4.9 Summary of grade 4 thrombocytopenia and platelets transfusions

| Patient | Total number of cycles received | Cycle numbers with grade 4 thrombocytopenia | Cycle numbers with platelets transfusions | Cycle numbers with dose reduction |
|---|---|---|---|---|

Listing 12.4.4.10 Summary of grade 4 anemia and EPO/transfusions

| Patient | Total number of cycles received | Cycle numbers with grade 4 anemia | Cycle numbers with EPO administration | i franchicióne | Cycle<br>numbers with<br>dose reduction |
|---|---|---|---|---|---|

Table 12.4.4.11 Platelet count time course pattern (summary)

| | | - | | se received | | | | |
|---|---|---|---|---|---|---|---|---|
| | 7 r | ng FD / 3.5 | 6 n | ng FD / 2.6<br>mg/m <sup>2</sup> | 5 1 | ng FD/2.0 | | Total |
| | | mg/m <sup>2</sup> | | mg/m² | mg/m <sup>2</sup> | | | |
| | N | Median | N | Median | N | Median | N | Median |
| | 11 | (range) | 11 | (range) | 11 | (range) | 1 4 | (range) |
| Platelet transfusion=Yes | | | | | | | | |
| Baseline grade 0 | | | | | | | | |
| | | 1 <sup>st</sup> cycle | | • | • | • | • | • |
| Onset day grade 4 | | | | | | | | |
| | 2 <sup>n</sup> | d cycle, 3rd cy | cle | | | | | |
| Onset day grade 4 | | | | | | | | |
| | | Total | | | | | | |
| Onset day grade 4 | | | | | | | | |
| Baseline grade 1, 2 | | | | | | | | |

| | | | Do | se received | | | | |
|---|---|---|---|---|---|---|---|---|
| | 7 n | ng FD / 3.5 | 6 n | ng FD / 2.6 | 5 r | ng FD/2.0 | | Total |
| | | mg/m <sup>2</sup> | | mg/m <sup>2</sup> | | mg/m <sup>2</sup> | | |
| | N | Median | N | Median | N | Median | N | Median |
| | | (range) | - ' | (range) | - ' | (range) | - ' | (range) |
| Platelet transfusion=No | | | | | | | | |
| Total | | | | | | | | |
| Total | | | | | | | | |
| | | 1 <sup>st</sup> cycle | | | | | | |
| Onset day grade 4 | | | | | | | | |
| | 2 <sup>n</sup> | d cycle, 3rd cy | cle | • | | | | |
| Onset day grade 4 | | | | | | | | |
| | | Total | | | | | | |
| Onset day grade 4 | | | | | | | | |
| Nadir day grade 4 | | | | | | | | |
| Nadir value grade 4 | | | | | | | | |
| Recovery day to grade ≤ 3 | | | | | | | | |
| Duration in days to grade 3 | | | | | | | | |
| Recovery day to grade ≤ 2 | | | | | | | | |
| Duration in days to grade 2 | | | | | | | | |
| Recovery day to grade ≤ 1 | | | | | | | | |
| Duration in days to grade 1 | | | | | | | | |

Table 12.4.4.12 Platelet count time course pattern (freqs)

| | | P | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | 7 n | ng FD / 3.5 | 6 m | g FD / 2.6<br>mg/m <sup>2</sup> | 5 r | ng FD/ 2.0<br>mg/m <sup>2</sup> | | Total |
| | | mg/m <sup>2</sup> | | mg/m <sup>2</sup> | | mg/m <sup>2</sup> | | |
| | N | % | N | % | N | % | N | % |
| Platelet transfusion=Yes | | | | | | | | |
| Baseline grade 0 | | | | | | | | |
| | | 1 <sup>st</sup> cycle | | | | | | |
| Onset day grade 4 | | | | | | | | |
| ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| | 2 <sup>n</sup> | d cycle, 3rd cy | cle | | | | | |
| Onset day grade 4 | | | | | | | | |
| ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| | | Total | | | | | | |
| Onset day grade 4 | | | | | | | | |
| ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| Baseline grade 1, 2 | | ı | | | | | | |
| Platelet transfusion=No | | | | | | | | |
| Total | | | | | | | | |
| Total | | | | | | | | |
| | | 1 <sup>st</sup> cycle | | | | | | |

| | | | Do | se received | | | | |
|---|---|---|---|---|---|---|---|---|
| | 7 n | ng FD / 3.5 | 6 n | ng FD / 2.6 | 5 t | ng FD/ 2.0 | | Total |
| | , 13 | $mg/m^2$ | 0 1 | $mg/m^2$ | | $mg/m^2$ | | |
| | N | % | N | % | N | % | N | % |
| Onset day grade 4 | | | | | | | | |
| ≤7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| | 2 <sup>n</sup> | cycle, 3 <sup>rd</sup> cy | cle | | l . | I | l . | |
| Onset day grade 4 | | | | | | | | |
| ≤7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| | | Total | | | | | | |
| Onset day grade 4 | | _ | | _ | | | | _ |
| ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| Nadir day grade 4 | | | | | | | | |
| ≤ 7<br>8-14 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| Recovery day to grade ≤ 3 | | | | | | | | |
| ≤ 22 | | | | | | | | |
| 23-28 | | | | | | | | |
| ≥ 29 | | | | | | | | |
| Duration in days to grade 3 | | | | | | | | |
| ≤ 5 | | | | | | | | |
| 6-10 | | | | | | | | |
| ≥11 | | | | | | | | |
| Recovery day to grade $\leq 2$ | | | | | | | | |
| ≤ 22 | | | | | | | | |
| 23-28 | | | | | | | | |
| ≥ 29 | | | | | | | | |
| Duration in days to grade 2 | | | | | | | | |
| ≤5 | | | | | | | | |
| 6-10 | | | | | | | | |
| ≥11 | | | | | | | | |
| Recovery day to grade ≤ 1 | | | | | | | | |
| ≤ 22 | | | | | | | | |
| 23-28 | | | | | | | | |
| ≥ 29 | | | | | | | | |
| Duration in days to grade 1 | | | | | | | | |
| ≤5 | | | | | | | | |
| 6-10 | | | | | | | | |
| ≥ 11 | | | | | | | | |

Table 12.4.4.13 Neutrophil count time course pattern (summary)

| 1 4010 12. 1. 1.15 1 (Cattopi | iii count timic | course par | | (Summary | , | | | |
|---|---|---|---|---|---|---|---|---|
| | | • | Do | se received | | | | |
| | 7 r | 7 mg FD / 3.5<br>mg/m <sup>2</sup> | | 6 mg FD / 2.6<br>mg/m <sup>2</sup> | | 5 mg FD/ 2.0<br>mg/m <sup>2</sup> | | Total |
| | N | Median<br>(range) | N | Median<br>(range) | N | Median<br>(range) | N | Median (range) |
| G-CSF=Yes | | | | | | | | |
| Baseline grade 0 | | | | | | | | |
| | | 1 <sup>st</sup> cycle | | | | | | |
| Onset day grade 4 | | | | | | | | |

| | 7 n | ng FD / 3.5 | 6 n | ng FD / 2.6 | 5 r | ng FD/ 2.0 | | Total |
|---|---|---|---|---|---|---|---|---|
| | | mg/m <sup>2</sup> | | mg/m <sup>2</sup> | | mg/m <sup>2</sup> | | |
| | N | Median | N | Median | N | Median | N | Median |
| | - ' | (range) | | (range) | - ' | (range) | - ' | (range) |
| | 2" | cycle, 3 <sup>rd</sup> cy | cle | • | | | | |
| Onset day grade 4 | | | | | | | | |
| | | Total | | | | | | |
| Onset day grade 4 | | | | | | | | |
| Baseline grade 1, 2 | | | 1 1 | | | | ı | |
| G-CSF=No | | | | | | | | |
| ••• | | | | | | | | |
| Total | | | | | | | | |
| Total | | . of | | | | | | |
| | | 1 <sup>st</sup> cycle | | | | | | |
| Onset day grade 4 | | | | | | | | |
| | | 1 4 4 7 | | | | | | |
| | 2" | cycle, 3rd cy | cle | • | | | | |
| Onset day grade 4 | | | | | | | | |
| | | Total | | | | | | |
| Onset day grade 4 | | | | | | | | |
| Nadir day grade 4 | | | | | | | | |
| Nadir value grade 4 | | | | | | | | |
| Recovery day to grade $\leq 3$ | | | | | | | | |
| Duration in days to grade 3 | | | | | | | | |
| Recovery day to grade $\leq 2$ | | | | | | | | |
| Duration in days to grade 2 | | | | | | | | |
| Recovery day to grade ≤ 1 | | | | | | | | |
| Duration in days to grade 1 | | | | | | | | |

Table 12.4.4.14 Neutrophil count time course pattern (freqs)

| • | | - | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | 7 r | ng FD / 3.5 | 6 r | ng FD / 2.6 | 5 ı | ng FD/ 2.0 | | Total |
| | | mg/m <sup>2</sup> | mg/m <sup>2</sup> | | | mg/m <sup>2</sup> | | |
| | N | % | N | % | N | % | N | % |
| G-CSF=Yes | | | | | | | | |
| Baseline grade 0 | | | | | | | | |
| | | 1 <sup>st</sup> cycle | | | | | | |
| Onset day grade 4 | | | | | | | | |
| ≤7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| | 2 <sup>n</sup> | d cycle, 3rd cy | cle | | | | | |
| Onset day grade 4 | | | | | | | | |
| ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| | | Total | | | | | | |
| Onset day grade 4 | | | | | | | | |
| ≤7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |

| | | | Do | se received | | | | |
|---|---|---|---|---|---|---|---|---|
| | 7 n | ng FD / 3.5 | | ng FD / 2.6 | 5 1 | ng FD/ 2.0 | 1 | Total |
| | | mg/m <sup>2</sup> | | mg/m <sup>2</sup> | | mg/m <sup>2</sup> | | |
| | N | % | N | % | N | % | N | % |
| Baseline grade 1, 2 | | | | | | | | |
| Baseline grade 1, 2 | | | | 1 | | 1 | | |
| G-CSF=N <sub>0</sub> | | | | | | | | |
| Total | | | | | | | | |
| Total | | | | | | | | |
| | | 1 <sup>st</sup> cycle | 1 | T | | T | | • |
| Onset day grade 4 | | | | | | | | |
| ≤7<br>8-14 | | | | | | | | |
| 8-14<br>≥ 15 | | | | | | | | |
| | 2 <sup>ne</sup> | cycle, 3 <sup>rd</sup> cy | cle | | 1 | ı | 1 | 1 |
| Onset day grade 4 | | | | | | | | |
| ≤7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| ··· | | Total | | | | | | |
| Onset day grade 4 | | Total | | | | | | |
| ≤7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| Nadir day grade 4 | | | | | | | | |
| ≤ 7<br>8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| Recovery day to grade $\leq 3$ | | | | | | | | |
| ≤ 22 | | | | | | | | |
| 23-28 | | | | | | | | |
| ≥ 29 | | | 1 | | | | | |
| Duration in days to grade 3 ≤ 5 | | | | | | | | |
| ≤ 3<br>6-10 | | | | | | | | |
| ≥ 11 | | | | | | | | |
| Recovery day to grade ≤ 2 | | | | | | | | |
| ≤ 22 | | | | | | | | |
| 23-28 | | | | | | | | |
| $\geq$ 29 Duration in days to grade 2 | | | | | | | | |
| ≤ 5 | | | | | | | | |
| 6-10 | | | | | | | | |
| ≥ 11 | | | | | | | | |
| Recovery day to grade ≤ 1 | | | | | | | | |
| ≤ 22 | | | | | | | | |
| 23-28<br>≥ 29 | | | | | | | | |
| Duration in days to grade 1 | | | <del> </del> | | | | 1 | |
| ≤ 5 | | | | | | | | |
| 6-10 | | | | | | | | |
| ≥ 11 | | | | | | | | |

Table 12.4.4.15 AST time course pattern (summary)

| There is in the first thing course p | accorn (summer) | |
|--------------------------------------|-----------------|-------|
| | Dose received | Total |

| | 7 n | ng FD / 3.5 | 6 n | ng FD / 2.6 | 5 ı | ng FD/2.0 | | |
|---|---|---|---|---|---|---|---|---|
| | | mg/m <sup>2</sup> | | mg/m <sup>2</sup> | | mg/m <sup>2</sup> | | |
| | N | Median<br>(range) | N | Median<br>(range) | N | Median<br>(range) | N | Median<br>(range) |
| Baseline grade 0 | | | | | | | | |
| | | 1 <sup>st</sup> cycle | | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| | 2 <sup>ne</sup> | cycle, 3rd cy | cle | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| | | Total | | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| Baseline grade 1, 2 | | | | | | | | |
| Total | | | | | | | | |
| | | 1 <sup>st</sup> cycle | | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| | 2 <sup>n</sup> | cycle, 3rd cy | cle | | | T | | |
| Onset day grade 3/4 | | | | | | | | |
| | | Total | | T | | T | | |
| Onset day grade 3/4 | | | | | | | | |
| Peak day grade 3/4 | | | | | | | | |
| Peak value grade 3/4 | | | | | | | | |
| Recovery day to grade ≤ 2 | | | | | | | | |
| Duration in days to grade 2 | | | | | | | | |
| Recovery day to grade ≤ 1 | | | | | | | | |
| Duration in days to grade 1 | | | | | | | | |

Table 12.4.4.16 AST time course pattern (freqs)

| | 7 mg FD / 3.5 mg/m² N % 1st cycle 2nd cycle, 3rd cy Total | | 6 m | ng FD / 2.6 | 5 r | ng FD/ 2.0 | | Total |
|---|---|---|---|---|---|---|---|---|
| | n | ng/m² | | mg/m <sup>2</sup> | mg/m <sup>2</sup> | | | |
| | | % | N | % | N | % | N | % |
| Baseline grade 0 | | | | | | | | |
| | | 1 <sup>st</sup> cycle | | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| | 2 <sup>nd</sup> ( | cycle, 3 <sup>rd</sup> cy | cle | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| | | Total | | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| Baseline grade 1, 2 | | | | • | | | | |

| | Dose received | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | 7 m | ng FD / 3.5 | 6 n | ng FD / 2.6 | 5 1 | ng FD/ 2.0 | | Total |
| | | mg/m <sup>2</sup> | | mg/m <sup>2</sup> | | mg/m <sup>2</sup> | | |
| | N | % | N | % | N | % | N | % |
| Total | | 1 <sup>st</sup> cycle | | | | | | |
| Onset day grade 3/4 | | 1 Cycle | 1 | | | | | |
| $\leq 7$ | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| | 2 <sup>nd</sup> | cycle, 3rd cy | cle | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| | | T 1 | | | | | | |
| Onset day grade 3/4 | 1 1 | Total | 1 | | 1 | I | | |
| Since the day grade 3/4 ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| Peak day grade 3/4 | | | | | | | | |
| ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| Recovery day to grade ≤ 2 | | | | | | | | |
| ≤22 | | | | | | | | |
| 23-28 | | | | | | | | |
| ≥ 29 | | | | | | | | |
| Duration in days to grade 2<br>≤ 5 | | | | | | | | |
| 6-10 | | | | | | | | |
| ≥ 11 | | | | | | | | |
| Recovery day to grade ≤ 1 | | | | | | | | |
| ≤22 | | | | | | | | |
| 23-28 | | | | | | | | |
| ≥ 29 | | | | | | | | |
| Duration in days to grade 1 | | | | | | | | |
| ≤5 | | | | | | | | |
| 6-10 | | | | | | | | |
| ≥11 | | | | | | | | |

Table 12.4.4.17 ALT time course pattern (summary)

| | | | | se received | | | | |
|---|---|---|---|---|---|---|---|---|
| | 7 n | ng FD / 3.5 | 6 mg FD / 2.6<br>mg/m <sup>2</sup> | | 5 mg FD/ 2.0<br>mg/m <sup>2</sup> | | | Total |
| | | | | mg/m <sup>2</sup> | $mg/m^2$ | | | |
| | N | Median (range) | N | Median (range) | N | Median (range) | N | Median (range) |
| Baseline grade 0 | | | | | | | | |
| | | 1 <sup>st</sup> cycle | | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| | 2 <sup>n</sup> | cycle, 3rd cy | cle | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| | | Total | | | | | | |
| Onset day grade 3/4 | | | | | | | | |

| | 7 n | ng FD / 3.5 | 6 n | 6 mg FD / 2.6 | | ng FD/2.0 | | Total |
|---|---|---|---|---|---|---|---|---|
| | | mg/m <sup>2</sup> | mg/m <sup>2</sup> | | mg/m <sup>2</sup> | | | |
| | N | Median<br>(range) | N | Median<br>(range) | N | Median (range) | N | Median (range) |
| Baseline grade 1, 2 | | | | | | | | |
| Total | | | | | | | | |
| | | 1 <sup>st</sup> cycle | | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| | 2 <sup>n</sup> | d cycle, 3rd cy | cle | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| | | Total | | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| Peak day grade 3/4 | | | | | | | | |
| Peak value grade 3/4 | | | | | | | | |
| Recovery day to grade $\leq 2$ | · | | | | · | | | |
| Duration in days to grade 2 | | | | | | | | |
| Recovery day to grade ≤ 1 | | | | | | | | |
| Duration in days to grade 1 | | | | | | | | |

Table 12.4.4.18 ALT time course pattern (freqs)

| 14010 12.1.1.10 1121 time e | | ( - 1-) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | 7 r | ng FD / 3.5 | | ng FD / 2.6 | 5 r | ng FD/ 2.0 | 1 | Total |
| | | $mg/m^2$ | | $mg/m^2$ | | $mg/m^2$ | | |
| | N | % | N | % | N | % | N | % |
| Baseline grade 0 | • | | | | | | | |
| <u> </u> | | 1 <sup>st</sup> cycle | | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| | 2 <sup>n</sup> | d cycle, 3rd cy | cle | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| | | Total | | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| ≤7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| Baseline grade 1, 2 | | | | | | • | | • |
| Total | | | | | | | | |
| | | 1 <sup>st</sup> cycle | | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| ≤7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| | 2 <sup>n</sup> | d cycle, 3rd cy | cle | • | | | | |
| Onset day grade 3/4 | | | | | | | | |
| ≤7 | | | | | | | | |
| 8-14 | | | | | | | | |

| | | | Do | se received | | | | |
|---|---|---|---|---|---|---|---|---|
| | 7 n | ng FD / 3.5 | 6 n | ng FD / 2.6 | 5 1 | ng FD/ 2.0 | | Total |
| | | mg/m <sup>2</sup> | | mg/m <sup>2</sup> | mg/m <sup>2</sup> | | | |
| | N | % | N | % | N | % | N | % |
| ≥ 15 | | | | | | | | |
| | | Total | | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| Peak day grade 3/4 | | | | | | | | |
| ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| Recovery day to grade $\leq 2$ | | | | | | | | |
| ≤ 22 | | | | | | | | |
| 23-28 | | | | | | | | |
| ≥ 29 | | | | | | | | |
| Duration in days to grade 2 | | | | | | | | |
| ≤5 | | | | | | | | |
| 6-10 | | | | | | | | |
| ≥ 11 | | | | | | | | |
| Recovery day to grade $\leq 1$ | | | | | | | | |
| ≤ 22 | | | | | | | | |
| 23-28 | | | | | | | | |
| ≥ 29 | | | | | | | | |
| Duration in days to grade 1 | | | | | | | | |
| ≤5 | | | | | | | | |
| 6-10 | | | | | | | | |
| ≥ 11 | | | | | | | | |

# 12.5 Physical Findings, PS, LVEF, ECG and Other Tests Related to Safety

# 12.5.1 Physical Findings and PS (ECOG)

Table 12.5.1.1 ECOG performance status during the study

| | | Cycle/PS* | | | | | |
|-------------|---|-----------|---|---|---|-----|-----|
| | 0 | 1 | 2 | 3 | 4 | ••• | EOT |
| Patient id. | | | | | | | |

<sup>(\*)</sup> Worst ECOG PS of the cycle determinations.

Table 12.5.1.2 Physical examination during the study

| | | Cycle/Physical examination result* | | | | |
|-------------|---|------------------------------------|---|---|---|-----|
| | 0 | 1 | 2 | 3 | 4 | EOT |
| Patient id. | | | | | | |

<sup>(\*)</sup> Worst result per cycle.

Table 12.5.1.3 Weight by patient per cycle

| | | Cycle/Weight |
|---|---|---|
| | 0<br>(kg) | $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ |
| Patient id. | | |

<sup>(\*) %</sup> of changes respect to baseline

## 12.5.2 LVEF, ECG and Other Related Tests

Listing 12.5.2.1 LVEF evolution during the study.

| Γ | | | LVEF(%) | |
|---|---------------|-----------|----------|-------------------|
| | Patient id. | LVEF(/0) | | |
| | 1 4010110 141 | Baseline* | Minimun* | End of treatment* |
| ſ | | | | |
| Ī | Median(Range) | | | |

<sup>(\*)</sup> LVEF (%) value and method

Listing 12.5.2.2 Electrocardiogram results. Evolution during the study.

| | | Cycle/ECG result* | | | | |
|-------------|---|-------------------|---|---|---|-----|
| | 0 | 1 | 2 | 3 | 4 | EOT |
| Patient id. | | | | | | |

<sup>(\*)</sup> Worst result of the cycle determinations.

Listing 12.5.2.3 Troponin I and Troponin T values. Evolution during the study.

| | | | | 2 |
|-------------|-------|------|-------|-----|
| Patient id. | Cycle | Test | Value | ULN |

# 12.6 Concomitant Therapy / Procedures According to the ATC Classification.

Table 12.6.1 Concomitant medication during treatment (ATC1, ATC2 and ATC4 levels)

| Concomitant medication at baseline | N | % |
|------------------------------------|---|---|
| Alimentary tract and metabolism | | |
| Antacids | | |
| Magnesium adipate | | |
| Blood and blood forming organs | | |
| Antithrombotic agents | | |
| Acenocoumarol | | |

Table 12.6.2 Summary of concomitant medication during treatment

| - | N | % |
|------------------------------------|---|---|
| No. of systems (ATC1 level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥ 3 | | |
| Median (range) | | |
| No. of indications (ATC2 level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥ 3 | | |
| Median (range) | | |
| No. of agent families (ATC4 level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥ 3 | | |
| Median (range) | | |
| No. of agents (PN level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥ 3 | | |
| Median (range) | | |

Listing 12.6.3 Patients with any transfusion during treatment

| U | | | J | | U | |
|---|---|---|---|---|---|---|
| Patient | Cycle | PM1183<br>dose in the<br>previous<br>cycle | Platelets /<br>RBC | Date first transfusion | Date last transfusion | No. of units required* |

<sup>(\*)</sup> No. of transfusions for platelets or no. of packed for RBC transfusions.

Listing 12.6.4 Patients with G-CSF during treatment

| _ | | | | | | | |
|---|---------|-------|-------|----|------|------------|----------|
| | Patient | Cycle | Agent | PT | Dose | Start date | End date |

# Table 12.6.5 Transfusions and G-CSF by dose

| | 7 mg FD | | $3.5 \text{ mg/m}^2$ | | Total | |
|--------------|---------|---|----------------------|---|-------|---|
| | N | % | N | % | N | % |
| Transfusions | | | | | | |
| RBC | | | | | | |
| Platelets | | | | | | |
| G-CSF | | | | | | |

Table 12.6.6 Subsequent therapy

| | N | % |
|--------------------------------------|---|---|
| Туре | | |
| Chemotherapy | | |
| Subsequent chemotherapy agents (ATC) | | |

Table 12.6.7 Subsequent therapy. Best response (if available).

| Tuble 12.0.7 Subsequent therapy. Best response (if available). | | | | | | |
|---|---|---|---|---|---|---|
| Best response | | Subsequent therapy | | | | |
| | | CR | PR | SD | PD | NE |
| PM01183 | CR | | | | | |
| | PR | | | | | |
| | SD | | | | | |
| | PD | | | | | |
| | NE | | | | | |

<sup>(\*)</sup> If a low number of best response to the subsequent therapy is available, a listing, instead of this table, will be provided.

#### APPENDIX II

# 13 DB Listings

#### CRF Listings.

- -Listing 13.1.1: Investigator comments
- -Listing 13.1.2: Study registration
- -Listing 13.1.3: Demography
- -Listing 13.1.4: Pregnancy test and adequate contraception
- -Listing 13.1.5: Prior medical history
- -Listing 13.1.6: Cancer history
- -Listing 13.1.7: Prior surgery
- -Listing 13.1.8: Prior radiotherapy
- -Listing 13.1.9: Prior medical therapy
- -Listing 13.1.10: Hematological laboratory values
- -Listing 13.1.11: Biochemical laboratory values
- -Listing 13.1.12: Coagulation laboratory values
- -Listing 13.1.13: Physical examination
- -Listing 13.1.14: Performance status
- -Listing 13.1.15: Vital signs
- -Listing 13.1.16: Electrocardiogram
- -Listing 13.1.17: LVEF
- -Listing 13.1.18: Prophylactic medication
- -Listing 13.1.19: Drug administration
- -Listing 13.1.20: Adverse events (including signs and symptoms)
- -Listing 13.1.21: Concomitant therapy/procedures
- -Listing 13.1.22: Tumor assessment
- -Listing 13.1.23: Evaluation of response by cycle
- -Listing 13.1.24: Best study overall response
- -Listing 13.1.25: End of treatment
- -Listing 13.1.26: Follow up
- -Listing 13.1.27: Death report form
- -Listing 13.1.28: Off study
- -Listing 13.1.29: BRCA 1/2 germline mutation

#### ICH Listings.

- -Listing 16.2.1 Discontinued patients
- -Listing 16.2.2 Protocol deviations
- -Listing 16.2.3 Patients excluded from the efficacy analysis
- -Listing 16.2.4 Demographic data
- -Listing 16.2.5 Compliance and-or Drug Concentration Data
- -Listing 16.2.6 Individual Efficacy Response data
- -Listing 16.2.7 Adverse event listings
- -Listing 16.2.8 Individual laboratory measurements

# 14 SAP Version History

#### 14.1 From version 1.0 to version 2.0

After the first version of the statistical plan was approved, some new protocol "substantial amendments No. 1 (Nov2013), No. 2 (Oct2014) and No. 3 (Feb2016)" were implemented. The Statistical Analysis Plan has been updated (changes are highlighted in *italic bold*) in accordance with the currently available version of the protocol (i.e., version 4) as follows:

### **Section 2 Study Design**

#### **Original text:**

This is a multicenter, open-label, exploratory, phase II clinical trial evaluating the efficacy and safety of PM01183 administration to patients with previously treated MBC, as follows.

Two Cohorts of MBC patients will be prospectively evaluated in the trial, initially according to germline BRCA1/2 status (mutated *vs.* unselected):

- Cohort A (BRCA+ Cohort): At least 53 evaluable patients with previously known deleterious BRCA1/2 mutation status at study entry.
- Cohort B (unselected Cohort): At least 64 evaluable patients without known deleterious BRCA1/2 mutation status at study entry, i.e., either:
  - o Patients known to have no deleterious BRCA1/2 mutations (BRCA-), or
  - Patients whose BRCA 1/2 mutation status is unknown (BRCA-UK);
     BRCA1/2 germline mutation status will be assessed in PM01183 responding patients in this subgroup.

[...]

An interim analysis based on the primary endpoint (ORR) is planned after 20 and 30 evaluable patients have been treated in Cohorts A and B, respectively (see Section  for details). If less than four out of 20 patients in Cohort A, or less than three out of 30 patients in Cohort B achieve an objective confirmed response, recruitment to that Cohort will be terminated.

### **Changed to:**

This is a multicenter, open-label, exploratory, phase II clinical trial evaluating the efficacy and safety of PM01183 administration to patients with previously treated MBC, as follows.

Two Cohorts of MBC patients will be prospectively evaluated in the trial according to germline BRCA1/2 status (mutated [Cohort A] vs. unselected [Cohort B]). A third Cohort (Cohort A1) will include advanced breast cancer patients with deleterious BRCA1/2 mutation status who received prior treatment with poly (ADP-ribose) polymerase (PARP) inhibitors:

- <u>Cohort A (BRCA+ Cohort)</u>: At least 53 evaluable patients with previously known deleterious BRCA1/2 mutation status at study entry.
- <u>Cohort A1 (BRCA+/PARPi Cohort):</u> 20 evaluable patients with known deleterious BRCA1/2 mutation status and prior treatment with PARP inhibitors (PARPi).
- <u>Cohort B (unselected Cohort)</u>: At least 64 evaluable patients without known deleterious BRCA1/2 mutation status at study entry, i.e., either:
  - o Patients known to have no deleterious BRCA1/2 mutations (BRCA-), or
  - Patients whose BRCA 1/2 mutation status is unknown (BRCA-UK); BRCA1/2 germline mutation status will be assessed in PM01183 responding patients in this subgroup.

[....]

An interim analysis based on the primary endpoint (ORR) is planned after 20 and 30 evaluable patients have been treated in Cohorts A and B, respectively (see Section  for details). No interim analysis is planned for Cohort A1. If less than four out of 20 patients in Cohort A, or less than three out of 30 patients in Cohort B achieve an objective confirmed response, recruitment to that Cohort will be terminated.

#### **Section 5.1 Sample Size**

#### **Original text**

The primary endpoint for this phase II study is to evaluate ORR.

- Cohort A (BRCA+): At least 53 evaluable patients will be recruited to test the null hypothesis that ORR is 20% or less (p ≤ 0.20) vs. the alternative hypothesis that 40% or more patients have objective response (p ≥ 0.4). With these assumptions, if the number of evaluable patients with objective response is ≥ 17, then this would allow the rejection of the null hypothesis.
- Cohort B (unselected): At least 64 evaluable patients will be recruited to test the null hypothesis that ORR is 10% or less ( $p \le 0.10$ ) vs. the alternative hypothesis that 25% or more patients have objective response ( $p \ge 0.25$ ). With these assumptions, if the number of evaluable patients with objective response is  $\ge 12$ , then this would allow the rejection of the null hypothesis.

The variance of the standardized tests is based on the null hypothesis. The type I error (alpha) associated with this one-sided test is 0.025 and the type II error (beta) is <0.1; hence, statistical power is > 90%. Futility analysis controlled by the Gamma family boundary will be performed when 20 and 30 patients have been evaluated in Cohorts A [Gm(-2)] and B [Gm(-1.5)], respectively. If less than four out of 20 patients in Cohort A, or less than three patients out of 30 in Cohort B achieve an objective response, recruitment to that Cohort will be stopped. Therefore, between 50 and at least 117 evaluable patients will be included in this study.

## Changed to:

The primary endpoint for this phase II study is to evaluate ORR.

#### Cohort A (BRCA+):

At least 53 evaluable patients will be recruited to test the null hypothesis that ORR is 20% or less ( $p \le 0.20$ ) vs. the alternative hypothesis that 40% or more patients have objective response ( $p \ge 0.4$ ). With these assumptions, if the number of evaluable patients with objective response is  $\ge 17$ , then this would allow the rejection of the null hypothesis.

#### • Cohort A1 (BRCA+/PARPi):

At least 20 evaluable patients will be included for an exploratory analysis: if the number of patients responding is  $\geq 4$  (20%), the lower limit of the exact binomial 95% confidence interval will be higher than 5% and thus lack of activity in this subpopulation will be ruled out.

## • Cohort B (unselected):

At least 64 evaluable patients will be recruited to test the null hypothesis that ORR is 10% or less ( $p \le 0.10$ ) vs. the alternative hypothesis that 25% or more patients have objective response ( $p \ge 0.25$ ). With these assumptions, if the number of evaluable patients with objective response is  $\ge 12$ , then this would allow the rejection of the null hypothesis.

The variance of the standardized tests is based on the null hypothesis. The type I error (alpha) associated with this one-sided test is 0.025 and the type II error (beta) is <0.1; hence, statistical power is >90%.

Futility analysis controlled by the Gamma family boundary will be performed when 20 and 30 patients have been evaluated in Cohorts A [Gm(-2)] and B [Gm(-1.5)], respectively. If less than four out of 20 patients in Cohort A, or less than three patients out of 30 in Cohort B achieve an objective response, recruitment to that Cohort will be stopped. Therefore, between 50 and at least 117 evaluable patients will be included in this study. About 110 evaluable patients are finally expected to be included in the three Cohorts: Cohort A (BRCA+), Cohort A1 (BRCA+/PARPi), and Cohort B (unselected).

#### **Section 6.2.2 Secondary Endpoints**

## **Original text:**

[...]

A log-rank test or Cox regression for time-to-event endpoints could be performed as supportive analysis to compare both Cohorts.

[...]

If appropriate, exploratory multivariate models (main effects or including interaction terms, if appropriate) will include all prognostic factors/covariates widely reported and recognized by oncologists: Cohort (BRCA (+) vs. BRCA (-) or unknown), BRCA (1 vs. 2 vs. both vs. negative/unkown), age, age at diagnosis, race (Caucasian vs. other), baseline Eastern Cooperative Oncology Group performance status (ECOG PS) (0 vs. >0), histology type (Ductal vs. lobular carcinoma), histology grade (poorly vs. other), stage at diagnosis,

primary tumor site (unilateral breast vs. bilateral), estrogen receptor (positive vs. negative), progesterone receptor (positive vs. negative), HER-2 receptor (positive vs. negative), site of current disease (CNS vs. liver vs. lung vs. non-visceral (including bone, skin, subcutaneous and lymph node) vs. other), liver metastases (yes vs. no), CNS metastases (yes vs. no), number of prior metastatic sites (1 vs. >1), body mass index (BMI), height, weight, body surface area (BSA), time from diagnosis to first infusion, prior surgery (yes vs. no), prior radiotherapy (yes vs. no), prior advanced treatment lines, prior advanced chemotherapy lines (1 vs. >1), prior anthracyclines (yes vs. no), prior taxane (yes vs. no), prior platinum (yes vs. no), anthracycline cumulative dose, last prior therapy PFS, first advanced chemotherapy PFS, last advanced chemotherapy PFS; PFS for anthracycline, taxane and platinum therapy, hormonotherapy (yes vs. no), adjuvant/neoadjuvant therapy (yes vs. no), presence of any bulky (< 50 mm vs. ≥ 50 mm) lesion, albumin at baseline, CA-15.3 or 27.29 at baseline, any relevant concomitant medication at baseline (to be determinate by the oncologist) (yes vs. no) and the sum of all target lesion diameters.

[...]

## **Changed to:**

[...]

A log-rank test or Cox regression for time-to-event endpoints could be performed as supportive analysis to compare both Cohorts between different cohorts and /or defined groups.

[...]

If appropriate, exploratory multivariate models (main effects or including interaction terms, if appropriate) will include all prognostic factors/covariates widely reported and recognized by oncologists: Cohort (BRCA (+) vs. BRCA (-) or unknown), BRCA (1 vs. 2 vs. both vs. negative/unkown), initial dose (7 mg FD vs 3.5 mg/m<sup>2</sup>), age, age at diagnosis, race (Caucasian vs. other), baseline Eastern Cooperative Oncology Group performance status (ECOG PS) (0 vs. >0), histology type (Ductal vs. lobular carcinoma), histology grade (poorly vs. other), stage at diagnosis, primary tumor site (unilateral breast vs. bilateral), hormone receptor positive (estrogen or progesterone receptor +, or both +) vs. triple negative, HER-2 receptor (positive vs. negative), site of current disease (CNS vs. liver vs. lung vs. non-visceral (including bone, skin, subcutaneous and lymph node) vs. other), liver metastases (yes vs. no), CNS metastases (yes vs. no), number of prior metastatic sites (1 vs. >1), body mass index (BMI), height, weight, body surface area (BSA), time from diagnosis to first infusion, prior surgery (ves vs. no), prior radiotherapy (ves vs. no), prior advanced treatment lines, prior advanced chemotherapy lines (0-1 vs. 2-3), prior anthracyclines (yes vs. no), prior taxane (yes vs. no), prior platinum (yes vs. no), prior PARPi (yes vs. no), anthracycline cumulative dose, last prior therapy PFS, first advanced chemotherapy PFS, last advanced chemotherapy PFS; PFS for anthracycline, taxane and platinum therapy, hormonotherapy (yes vs no), adjuvant/neoadjuvant therapy (yes vs no), presence of any bulky ( $< 50 \text{ mm } vs. \ge 50 \text{ mm}$ ) lesion, albumin at baseline, CA-15.3 or 27.29 at baseline, any relevant concomitant medication at baseline (to be determinate by the oncologist) (yes vs. no) and the sum of all target lesion diameters.

## **Section 8.9 Subgroup Analysis**

## **Original Text:**

The analysis will be done by Cohort and additionally, if clinically appropriate, the two Cohorts might be pooled into one, whenever differences between Cohorts are considered not relevant. In such case, the point estimates and their 95% CIs will be also reassessed in order to obtain more accurate calculations.

No other specific subgroup analysis is being planned for the analysis. However, if any of the disease characteristics is sufficiently represented and clinically relevant, subgroup analysis may be performed in order to explore the activity of PM01183 in specific breast cancer subpopulations according to hormonal receptor status, HER-2 overexpression, number and/or type of prior therapies, or according to other available histological/molecular classifications.

#### Changed to:

The analysis will be done by Cohort and additionally, if clinically appropriate, the two Cohorts might be pooled into one, whenever differences between Cohorts are considered not relevant. In such case, the point estimates and their 95% CIs will be also reassessed in order to obtain more accurate calculations.

Efficacy subgroup analysis will be performed in Cohort A according to prior treatment with platinum, BRCA status (BRCA1 vs. BRCA2), hormonal status (Triple negative vs HR+), number of advanced chemotherapy lines (0-1 vs. 2-3) and starting dose (7 mg FD vs. 3.5 mg/m<sup>2</sup>).

Safety subgroup analysis will be performed according to starting dose (7 mg FD vs. 3.5  $mg/m^2$ ), these analysis include laboratory abnormalities and adverse events.

No other specific subgroup analysis is being planned for the analysis. However, if any of the disease characteristics is sufficiently represented and clinically relevant, If clinically relevant, other subgroup analysis may be performed in order to explore the activity of PM01183 in specific breast cancer subpopulations. according to hormonal receptor status, HER-2 overexpression, number and/or type of prior therapies, or according to other available histological/molecular classifications.
#### **Section 11.3 Efficacy Analysis**

#### **Original text:**

Efficacy analysis will be carried out on the "All Evaluable Patients" population.

If any of the disease characteristics is sufficiently represented and clinically relevant, subgroup analysis may be performed in order to explore the activity of PM01183 in specific breast cancer subpopulations according to hormonal receptor status, HER-2 overexpression, number and/or type of prior therapies, or according to other available histological/molecular classifications.

#### Changed to:

Efficacy analysis will be carried out on the "All Evaluable Patients" population.

Subgroup analysis will be performed in Cohort A according to prior treatment with platinum, BRCA status (BRCA1 vs. BRCA2), hormonal status (Triple negative vs. HR+), number of advanced chemotherapy lines (0-1 vs. 2-3) and starting dose (7 mg FD vs. 3.5 mg/m²).

The tables included in each subgroup analysis are the following:

Table 11.3.1.1 Response rate

Table 11.3.1.2 Overall response rate

Table 11.3.2.1 Duration of response

Table 11.3.2.2 Progression-free survival (PFS)

Table 11.3.2.3 Overall survival (OS)

The tables will be annotated by adding a letter as suffix:

- BRCA status: a
- Prior platinum: b
- Hormonal status: c
- Advanced chemotherapy lines: d
- Starting dose: e

If any of the other disease characteristics is sufficiently represented and clinically relevant, subgroup analysis may be performed, and their corresponding tables will also be annotated by adding a letter to the table's name. according to hormonal receptor status, HER-2 overexpression, number and/or type of prior therapies, or according to other available histological/molecular classifications.

#### **Section 12.1 Extent of Exposure**

#### Added text:

Subgroup analysis will be performed according to starting dose (7 mg FD vs. 3.5 mg/m<sup>2</sup>). The tables will be annotated by adding a letter as suffix.

The tables included in the subgroup analysis are the following:

Table 12.1.1.1 Number of cycles administered and dose intensity

Table 12.1.2.1.3 Number of patients and cycles with dosing delay according to relationship

Table 12.1.3.3 Number of patient and cycles with dose reduction according to relationship

#### **Section 12.2.1 Adverse Events**

#### Added text:

Subgroup analysis will be performed according to starting dose (7 mg FD vs. 3.5 mg/m²) and Cohort.

The groups will include:

- Patient treated at 7 mg FD Cohort B
- Patient treated at 7 mg FD Cohort A
- Patient treated at 7 mg FD any Cohort
- Patient treated at 3.5 mg/m<sup>2</sup> Cohort A
- Patient treated at 3.5 mg/m<sup>2</sup> Cohort A1
- Patient treated at 3.5 mg/m<sup>2</sup> any Cohort

The tables will be annotated by adding a letter as suffix.

The tables included in the subgroup analysis are the following:

Table 12.2.2.2 Treatment related AEs. Worst grade by patient

Table 12.2.2.3 Treatment related AEs. Worst grade by cycle

Table 12.2.2.4 Adverse events regardless of relationship. Worst grade by patient

Table 12.2.2.5 Adverse events regardless of relationship. Worst grade by cycle

## **Section 12.4 Clinical Laboratory Evaluation**

#### Added text:

Subgroup analysis will be performed according to starting dose (7 mg FD vs. 3.5 mg/m²) and Cohort.

The groups will include:

- Patient treated at 7 mg FD Cohort B
- Patient treated at 7 mg FD Cohort A
- Patient treated at 7 mg FD any Cohort
- Patient treated at 3.5 mg/m<sup>2</sup> Cohort A
- Patient treated at 3.5 mg/m<sup>2</sup> Cohort A1
- Patient treated at 3.5 mg/m<sup>2</sup> any Cohort

The tables will be annotated by adding a letter as suffix.

The tables included in the subgroup analysis are the following:

Table 12.4.1.1 Hematological abnormalities during treatment, worst grade per patient

Table 12.4.1.2 Hematological abnormalities during treatment, worst grade per cycle

Table 12.4.2.1 Biochemical abnormalities during treatment, worst grade per patient

Table 12.4.2.2 Biochemical abnormalities during treatment, worst grade per cycle

Table 12.4.3.1 Coagulation abnormalities during treatment, worst grade per patient

Table 12.4.3.2 Coagulation abnormalities during treatment, worst grade per cycle

#### 14.2 From version 2.0 to version 3.0

The Statistical Analysis Plan has been updated (changes are highlighted in *italic bold*) in order to include some relevant analysis according to the medical responsible, to clarify some of the analyses and to correct several typos found in the previous SAP version.

#### **Section 5.1 Sample size**

#### **Original text:**

[...]

#### Cohort A1 (BRCA+/PARPi):

At least 20 evaluable patients will be for an exploratory analysis: if the number of patients responding is  $\geq$  4 (20%), the lower limit of the exact binomial 95% confidence interval will be higher than 5% and thus lack of activity in this subpopulation will be ruled out.

#### **Changed to:**

[...]

#### • Cohort A1 (BRCA+/PARPi):

At least 20 evaluable patients will be *recruited* for an exploratory analysis: if the number of patients responding is  $\geq$  4 (20%), the lower limit of the exact binomial 95% confidence interval will be higher than 5% and thus lack of activity in this

#### **Section 6.2.2 Secondary Endpoints**

#### **Original text:**

[...]

If relevant, efficacy parameters versus baseline covariates will be analyzed and appropriate test will be used (i.e., the Fisher exact test and logistic regression for categorical variables, the log-rank test or Cox regression for time-to-event variables, etc.).

If appropriate, exploratory multivariate models (main effects or including interaction terms, if appropriate) will include all prognostic factors/covariates widely reported and recognized by oncologists: Cohort (BRCA (+) vs. BRCA (-) or unknown), BRCA (1 vs. 2 vs. both vs. negative/unkown), initial dose (7 mg FD vs 3.5 mg/m<sup>2</sup>), age, age at diagnosis, race (Caucasian vs. other), baseline Eastern Cooperative Oncology Group performance status (ECOG PS) (0 vs. >0), histology type (Ductal vs. lobular carcinoma), histology grade (poorly vs. other), stage at diagnosis, primary tumor site (unilateral breast vs. bilateral), hormone receptor positive (estrogen or progesterone receptor +, or both +) vs. triple negative, HER-2 receptor (positive vs. negative), site of current disease (CNS vs. liver vs. lung vs. non-visceral (including bone, skin, subcutaneous and lymph node) vs. other), liver metastases (yes vs. no), CNS metastases (yes vs. no), number of prior metastatic sites (1 vs. >1), body mass index (BMI), height, weight, body surface area (BSA), time from diagnosis to first infusion, prior surgery (yes vs. no), prior radiotherapy (yes vs. no), prior advanced treatment lines, prior advanced chemotherapy lines (0-1 vs. 2-3), prior anthracyclines (ves vs. no), prior taxane (yes vs. no), prior platinum (yes vs. no), prior PARPi (yes vs. no), anthracycline cumulative dose, last prior therapy PFS, first advanced chemotherapy PFS, last advanced chemotherapy PFS; PFS for anthracycline, taxane and platinum therapy, hormonotherapy (yes vs no), adjuvant/neoadjuvant therapy (yes vs no), presence of any bulky ( $< 50 \text{ mm vs.} \ge 50 \text{ mm}$ ) lesion, albumin at baseline, CA-15.3 or 27.29 at baseline, any relevant concomitant medication at baseline (to be determinate by the oncologist) (ves vs. no) and the sum of all target lesion diameters.

All variables with a good percentage of valid cases (approximately  $\geq 90\%$ ) will be included in the exploratory multivariate analysis. [...]

### Changed to:

[...]

If appropriate, exploratory multivariate models (main effects or including interaction terms, if appropriate) will include all prognostic factors/covariates widely reported and recognized by oncologists: Cohort (BRCA (+) vs. BRCA (-) or unknown), BRCA (1 vs. 2 vs. both vs. negative/unknown in cohorts A and A1), initial dose (7 mg FD vs 3.5 mg/m²), age, age at diagnosis, race (Caucasian vs. other), baseline Eastern Cooperative Oncology Group performance status (ECOG PS) (0 vs. >0), histology type (Ductal vs. lobular carcinoma), histology grade (poorly vs. other), stage at diagnosis, primary tumor site (unilateral breast vs. bilateral), hormone receptor positive (estrogen or progesterone receptor +, or both +)

vs. triple negative, HER-2 receptor (positive vs. negative), site of current disease *such as liver metastases (yes vs. no), CNS metastases (yes vs. no), lung metastases (yes vs. no), (CNS vs. liver vs.* non-visceral (including bone, skin, subcutaneous and lymph node) vs. other), *liver metastases (yes vs. no), CNS metastases (yes vs. no),* number of prior metastatic sites (1 vs. >1), body mass index (BMI), height, weight, body surface area (BSA), time from diagnosis to first infusion, prior surgery (yes vs. no), prior radiotherapy (yes vs. no), prior advanced treatment lines, prior advanced chemotherapy lines (0-1 vs. 2-3), prior anthracyclines (yes vs. no), prior taxane (yes vs. no), prior platinum (yes vs. no), prior PARPi (yes vs. no), *anthracycline cumulative dose*, last prior therapy PFS, first advanced chemotherapy PFS, last advanced chemotherapy PFS, PFS for anthracycline, taxane and platinum therapy, hormonotherapy (yes vs no), adjuvant/neoadjuvant therapy (yes vs no), *platinum-free interval (in months)*, presence of any bulky (< 50 mm vs. ≥ 50 mm) lesion, albumin at baseline, CA-15.3 or 27.29 at baseline, any relevant concomitant medication at baseline (to be determinate by the oncologist) (yes vs. no) and the sum of all target lesion diameters.

All variables with a good percentage of valid cases (approximately  $\geq 90\%$ ) and with a p-value lower than 0.10 in the univariate analysis will be included in the exploratory multivariate analysis. [...]

If appropriate, multivariate analysis will be produced for a relevant subgroup of patients (e.g. by cohort).

#### **Section 8.3 Baseline and Demographic Data**

#### Original text

[...]

In case of pre-treatment characteristics with multiple measurements per subject before the start of treatment (laboratory assessments, vital signs) the baseline measurement will be considered the last value prior to or on the first day of treatment.

## **Changed to:**

[...]

In case of pre-treatment characteristics with multiple measurements per subject before the start of treatment (laboratory assessments, vital signs) the baseline measurement will be considered the last value prior to or on the first day of treatment.

Baseline and demography characteristics in different subgroups of analysis (i.e. cohorts) will be compared by means of Fisher's exact test (categorical variables) and Mann-Whitney-Wilcoxon (continuous variables).

#### **Section 8.8 Imputation of incomplete dates**

#### Added:

Between treatment start and end of treatment

All date variables during treatment where information is needed and is not fully available, for example adverse events or concomitant medications, will be subject of imputation by means of SAS programming. If the day of a date is unknown then the imputed day will be 1, if the month and/or year is also unknown then the imputed date will 1/January (this assumption will be valid if the imputed date is not earlier than the treatment start date; otherwise, the imputed date will be the treatment start date).

#### **Section 8.9 Subgroup Analysis**

### **Original text:**

[...]

Efficacy subgroup analysis will be performed in Cohort A according to prior treatment with platinum (Yes Vs No), BRCA status (BRCA1 vs. BRCA2), hormonal status (Triple negative vs. HR+), number of advanced chemotherapy lines (0-1 vs. 2-3) and starting dose (7 mg FD vs. 3.5 mg/m²).

#### Changed to:

[...]

Efficacy subgroup analysis will be performed in Cohort A according to prior treatment with platinum (Yes vs. 4/s No), BRCA status (BRCA1 vs. BRCA2), hormonal status (Triple negative vs. HR+), number of advanced chemotherapy lines (0-1 vs. 2-3), prior PARPi (Yes vs. No) and starting dose (7 mg FD vs. 3.5 mg/m²).

Additional efficacy subgroup analysis will be performed in Cohorts A+A1 according to prior PARPi (Yes vs. No).

#### Table 11.1.4.3 Number of lines of prior therapy

**Typo correction:** Antracycline has been corrected to Anthracycline.

#### Table 11.1.6.3 Baseline characteristics: Electrocardiogram values

**Original table:** 

| - 8 | | | | |
|--------------------|---|--------|-----|-----|
| Parameter | N | Median | Min | Max |
| PR interval (msec) | | | | |
| Heart rate (bpm) | | | | |
| QT interval (msec) | | | | |
| QRS complex (msec) | | | | |
| QTc Bazett's* | | | | |

<sup>(\*)</sup> QTc (Bazett's) = QT interval /  $\sqrt{(60/\text{Heart rate})}$ 

| Parameter | N | Median | Min | Max |
|--------------------------|---|--------|-----|-----|
| PR interval (msec) | | | | |
| Heart rate (bpm) | | | | |
| QT interval (msec) | | | | |
| QRS complex (msec) | | | | |
| QTc Fridericia Bazett's* | | | | |

## Listing 11.1.6.4 Patients with abnormal electrocardiogram

**Original listing:** 

| Patient id. | Abnormality | Details* | Reason for<br>clinically<br>indicated<br>repeat | PR interval (msec) | Heart rate (bpm) | QT interval (msec) | QRS<br>complex<br>(msec) | QTc<br>Bazett's** |
|---|---|---|---|---|---|---|---|---|

<sup>(\*)</sup>For non-significant abnormalities, for further details see prior medical history or Signs and symptoms; (\*\*) QTc (Bazett's) = QT interval /  $\sqrt{(60/\text{Heart rate})}$ 

**Changed to:** 

| Patient id. | Abnormality | Details* | Reason for<br>clinically<br>indicated<br>repeat | PR<br>interval<br>(msec) | Heart rate (bpm) | QT<br>interval<br>(msec) | QRS<br>complex<br>(msec) | QTc<br>Fridericia <i>Bazett's</i> ** |
|---|---|---|---|---|---|---|---|---|

<sup>(\*)</sup>For non-significant abnormalities, for further details see prior medical history or Signs and symptoms;  $\frac{(**)}{QTe}$  (Bazett's) =  $\frac{QT}{QT}$  interval  $\frac{1}{\sqrt{(60/Heart rate)}}$ 

## Listing 11.1.10.4 Signs and Symptoms at baseline

**Original listing:** 

| Patient id. | Sign/symptom | Grade* | Onset date | Relationship | Treated* |
|-------------|--------------|--------|------------|--------------|----------|

Changed to:

| Patient id. | Sign/symptom | Grade* | Onset date | Relationship | <del>Treated*</del> |
|---|---|---|---|---|---|

## Section 11.1.12 Baseline and demographic characteristic comparisons

#### **Section added:**

Table 11.1.12.1 Baseline and demographic characteristic comparisons by cohorts

| | | N | Cohort A | Cohort A1 | Cohort B | p-value* |
|---|---|---|---|---|---|---|
| Age | Median (range) | X | X.X (XX-XX) | X.X (XX-XX) | X.X (XX-XX) | X.XXXX |
| PS (ECOG) | 0 | X | X ( XX.X %) | X ( XX.X %) | X ( XX.X %) | X.XXXX |
| | 1 | • | X ( XX.X %) | X ( XX.X %) | X ( XX.X %) | |
| BSA | Median (range) | | | | | |
| BRCA mutation | 1 | | | | | |
| | 2 | | | | | |
| Receptor status | Triple negative | | | | | |
| | HR+/HER2 - | | | | | |

| | | N | Cohort A | Cohort A1 | Cohort B | p-value* |
|---|---|---|---|---|---|---|
| | HER2 + | | | | | |
| Liver metastases | Yes | | | | | |
| | No | | | | | |
| CNS metastases | Yes | | | | | |
| | No | | | | | |
| Sites involvement | <3 sites | | | | | |
| | ≥3 sites | | | | | |
| Advanced lines | Median (range) | | | | | |
| Advanced CT lines | Median (range) | | | | | |
| Prior Platinum | Yes | | | | | |
| | No | | | | | |
| Prior Anthracyclines | Yes | | | | | |
| | No | | | | | |
| Prior Taxanes | Yes | | | | | |
| | No | | | | | |
| Prior Capecitabine | Yes | | | | | |
| | No | | | | | |
| Prior PARP Inhibitor | Yes | | | | | |
| | No | | | | | |

<sup>\*</sup>Fisher's exact test (categorical variables); Mann-Whitney-Wilcoxon (continuous variables)

Table 11.1.12.2 Baseline and demographic characteristic comparisons: Platinum Yes/No in Cohort A

| | | | Prior platinum | Prior platinum | |
|-----------|----------------|---|----------------|----------------|----------|
| | | N | Yes | No | p-value* |
| Age | Median (range) | X | X.X (XX-XX) | X.X (XX-XX) | X.XXXX |
| PS (ECOG) | 0 | X | X ( XX.X %) | X ( XX.X %) | X.XXXX |
| | 1 | | X ( XX.X %) | X ( XX.X %) | |
| | ••• | | | | |

<sup>\*</sup>Fisher's exact test (categorical variables);Mann-Whitney-Wilcoxon (continuous variables). For the complete list of covarites, see table 11.1.12.1

Table 11.1.12.3 Baseline and demographic characteristic comparisons: BRCA 1 vs 2 in Cohort A

| | | N | BRCA 1 | BRCA 2 | p-value* |
|-----------|----------------|---|-------------|-------------|----------|
| Age | Median (range) | X | X.X (XX-XX) | X.X (XX-XX) | X.XXXX |
| PS (ECOG) | 0 | X | X ( XX.X %) | X ( XX.X %) | X.XXXX |

| | N | BRCA 1 | BRCA 2 | p-value* |
|---|---|-------------|-------------|----------|
| 1 | • | X ( XX.X %) | X ( XX.X %) | |

<sup>\*</sup>Fisher's exact test (categorical variables); Mann-Whitney-Wilcoxon (continuous variables). For the complete list of covarites, see table 11.1.12.1

Table 11.1.12.4 Baseline and demographic characteristic comparisons: Prior PARPi Yes/No in Cohorts A+A1

| 100/110 | th Contorts 11 -111 | | | | |
|---|---|---|---|---|---|
| | | N | Prior PARPi<br>Yes | Prior PARPi<br>No | p-value* |
| Age | Median (range) | X | X.X (XX-XX) | X.X (XX-XX) | X.XXXX |
| PS (ECOG) | 0 | X | X ( XX.X %) | X ( XX.X %) | X.XXXX |
| | 1 | | X ( XX.X %) | X ( XX.X %) | |

<sup>\*</sup>Fisher's exact test (categorical variables); Mann-Whitney-Wilcoxon (continuous variables). For the complete list of covarites, see table 11.1.12.1

Table 11.1.12.5 Baseline and demographic characteristic comparisons: Initial dose 7 mg FD vs 3.5 mg/m<sup>2</sup> in Cohort A

| | | N | 7 mg FD | $3.5 \text{ mg/m}^2$ | p-value* |
|---|---|---|---|---|---|
| Age | Median (range) | X | X.X (XX-XX) | X.X (XX-XX) | X.XXXX |
| PS (ECOG) | 0 | X | X ( XX.X %) | X ( XX.X %) | X.XXXX |
| | 1 | • | X ( XX.X %) | X ( XX.X %) | |
| | ••• | | | | |

<sup>\*</sup>Fisher's exact test (categorical variables); Mann-Whitney-Wilcoxon (continuous variables). For the complete list of covarites, see table 11.1.12.1

Table 11.1.12.6 Baseline and demographic characteristic comparisons: Hormonal status triple negative vs Other

| | | N | Triple negative<br>Yes | Triple negative | p-value* |
|---|---|---|---|---|---|
| Age | Median (range) | X | X.X (XX-XX) | X.X (XX-XX) | X.XXXX |
| PS (ECOG) | 0 | X | X ( XX.X %) | X ( XX.X %) | X.XXXX |
| | 1 | | X ( XX.X %) | X ( XX.X %) | |
| | ••• | | | | |

<sup>\*</sup>Fisher's exact test (categorical variables);Mann-Whitney-Wilcoxon (continuous variables). For the complete list of covarites, see table 11.1.12.1

Table 11.1.12.7 Baseline and demographic characteristic comparisons: Advanced chemotherapy lines

| | | N | 0-1 lines | >1 lines | p-value* |
|-----------|----------------|---|-------------|-------------|----------|
| Age | Median (range) | X | X.X (XX-XX) | X.X (XX-XX) | X.XXXX |
| PS (ECOG) | 0 | X | X ( XX.X %) | X ( XX.X %) | X.XXXX |
| | 1 | | X ( XX.X %) | X ( XX.X %) | |

<sup>\*</sup>Fisher's exact test (categorical variables);Mann-Whitney-Wilcoxon (continuous variables). For the complete list of covarites, see table 11.1.12.1

#### **Section 11.3 Efficacy Analysis**

#### **Original text:**

Efficacy analysis will be carried out on the "All Evaluable Patients" population.

Subgroup analysis will be performed in Cohort A according to prior treatment with platinum, BRCA status (BRCA1 vs. BRCA2), hormonal status (Triple negative vs. HR+), number of advanced chemotherapy lines (0-1 vs. 2-3) and starting dose (7 mg FD vs. 3.5 mg/m²).

The tables included in each subgroup analysis are the following:

[...]

- Prior PARPi: f

#### Changed to:

Efficacy analysis will be carried out on the "All Evaluable Patients" population.

Subgroup analysis will be performed in Cohort A according to prior treatment with platinum, BRCA status (BRCA1 vs. BRCA2), hormonal status (Triple negative vs. HR+), number of advanced chemotherapy lines (0-1 vs. 2-3), prior PARPi (Yes vs. No) and starting dose (7 mg FD vs. 3.5 mg/m<sup>2</sup>).

Subgroup analysis will be performed in Cohorts A+A1 according to prior PARPi (Yes vs. No).

The tables included in each subgroup analysis are the following:

[...]

- Prior PARPi (Cohort A): f
- Prior PARPi (Cohorts A+A1): g

Listing 11.3.2.5 Characteristics of patients with clinical benefit\*

**Original listing:** 

| Oligina | | 8 | Histologo | Hormonal<br>Status<br>(ER +/-; PR | No.<br>of<br>prior | No. of advanced prior lines | I | Prior last thera | пру |
|---|---|---|---|---|---|---|---|---|---|
| Patient | PS /<br>Age | Histology<br>Type | Histology<br>Grade | +/-; HER2<br>+/-) | lines | prior miles | Agents | Best<br>response | PFS (months) |

| Patient | Cycles received | Best response | PFS (months) | OS<br>(months) | DR (months) |
|---|---|---|---|---|---|

**Changed to:** 

| | 5 ca c | • | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Hormonal<br>Status<br>(ER +/-;<br>PR +/-; | | No.<br>of<br>prior<br>lines | No. of advanced <i>CT prior</i> lines | Prior<br>Platinum<br>(Y/N) | Best<br>response<br>Prior<br>platinum | | Prior last therapy | |
| Patient | PS / | BRCA | Histology | Histology | HER2 +/- | Sites | | | | _ | Agents | Best<br>response | PFS<br>(month |
| | Age | status | Type | Grade | , | | | | | | | | |

| Patient | Initial dose | Cycles received | Best response | PFS (months) | OS<br>(months) | DR (months) |
|---|---|---|---|---|---|---|

## Section 11.3.2 Secondary analyses

#### Added:

Figure 11.3.2.8 "Swimmer plot" PFS in Cohort A



Figure 11.3.2.9 "Swimmer plot" PFS in Cohort A1



Figure 11.3.2.10 "Swimmer plot" PFS in Cohort B



## **Section 11.3.3 Exploratory Multivariate Analysis**

Section title has been modified.

## **Original title:**

11.3.3 Exploratory Multivariate Analysis

## **Changed to:**

11.3.3 Exploratory *Univariate and* Multivariate Analyses

## **Original section:**

Table 11.3.3.1 Multivariate analysis of response rate

| | Analysis of Maximum Likelihood Estimates |
|---|---|
| Variable label Variable values DF Estimate Standard error Wald chisquare Pr > ChiSq Odds ratio estimate 95% Vocnfid lim | |

(See list of covariates in section 6.2.2).

Table 11.3.3.2 Multivariate analysis of PFS

| | 4010 11.5.5.2 Wildie Variate analysis of 115 |
|---|---|
| | Analysis of Maximum Likelihood Estimates |
| Variable label Variable values DF Parameter estimate error Chi-square Pr > ChiSq Hazard ratio confideration limits | |

| | Analysis of Maximum Likelihood Estimates |
|---|---|
| Variable label Variable values DF Parameter estimate Chi-square Pr > ChiSq Hazard ratio confidence of the confidence of | |

(See list of covariates in section 6.2.2).

Table 11.3.3.3 Multivariate analysis of OS

| | doto 11.5.5.5 Whater whateful of OB |
|---|---|
| | Analysis of Maximum Likelihood Estimates |
| Variable label Variable values DF Parameter estimate Chi-square Pr > ChiSq Hazard 95% Hazard ratio confidence ratio limits | |

(See list of covariates in section 6.2.2).

## Changed to:

Table 11.3.3.1 Univariate analysis of response rate

| Variable<br>label | Variable<br>values | DF | Estimate | Standard<br>error | Wald chi-<br>square | Pr > ChiSq | Odds ratio<br>estimate | 95% Odds<br>Ratio<br>confidence<br>limits |
|---|---|---|---|---|---|---|---|---|

(See list of covariates in section 6.2.2).

Table 11.3.3.1 11.3.3.2 Multivariate analysis of response rate

| Analysis of Maximum Likelihood Estimates | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable label | Variable<br>values | DF | Estimate | Standard<br>error | Wald chi-<br>square | Pr > ChiSq | Odds ratio estimate | 95% <i>Wald Odds Ratio</i> confidence limits |

(See list of covariates in section 6.2.2. Only those covariates with a p-value < 0.10 in univariate analysis and with a 90% of valid observations will be included).

Table 11.3.3.3 Univariate analysis of PFS

| Variable<br>label | Variable<br>values | DF | Parameter<br>estimate | Standard<br>error | Chi-<br>square | Pr > ChiSq | Hazard<br>ratio | 95% Hazard ratio<br>confidence<br>limits |
|---|---|---|---|---|---|---|---|---|

(See list of covariates in section 6.2.2).

Table 11.3.3.2 11.3.3.4 Multivariate analysis of PFS

Analysis of Maximum Likelihood Estimates

| Variable label | Variable values | DF | Parameter estimate | Standard<br>error | Chi-square | Pr > ChiSq | Hazard<br>ratio | 95% Hazard ratio confidence limits |
|---|---|---|---|---|---|---|---|---|

(See list of covariates in section 6.2.2. Only those covariates with a p-value < 0.10 in univariate analysis and with a 90% of valid observations will be included).

Table 11.3.3.5 Univariate analysis of OS

| Variable<br>label | Variable<br>values | DF | Parameter<br>estimate | Standard<br>error | Chi-<br>square | Pr > ChiSq | Hazard<br>ratio | 95% Hazard ratio<br>confidence<br>limits |
|---|---|---|---|---|---|---|---|---|

(See list of covariates in section 6.2.2).

Table 11.3.3.3 11.3.3.6 Multivariate analysis of OS

| | adole 11.0.0.0 11.0.0.0 11.0.0.0 11.0.0.0 11.0.0.0 01.0.0 | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Analysis of Maximum Likelihood Estimates | | | | | | | | |
| Variable label | Variable values | DF | Parameter estimate | Standard<br>error | Chi-square | Pr > ChiSq | Hazard ratio | 95% Hazard ratio confidence limits |

(See list of covariates in section 6.2.2. Only those covariates with a p-value < 0.10 in univariate analysis and with a 90% of valid observations will be included).

## Table 12.1.2.1.2 Number of patients and cycles with dosing delay, any relationship

**Original table:** 

| | N | % |
|------------------------------------------|---|---|
| No. of patients treated | | |
| No. of patients with any dose delay | | |
| No. of cycles administered | | |
| No. of cycles susceptible to be delayed* | | |
| No. of cycles with dosing delay** | | |
| No. of patients with | | |
| No cycles delayed | | |
| 1 cycle delayed | | |
| 2 cycles delayed | | |
| ≥ 3 cycles delayed | | |

| | N | % |
|------------------------------------------------------|---|---|
| No. of patients treated | | |
| No. of patients susceptible to have any dose delayed | | |
| No. of patients with any dose delayed | | |
| No. of cycles administered | | |
| No. of cycles susceptible to be delayed* | | |
| No. of cycles with dosing delay** | | |
| No. of patients with | | |
| No cycles delayed | | |
| 1 cycle delayed | | |
| 2 cycles delayed | | |
| ≥ 3 cycles delayed | | |

# Table 12.1.2.1.4 Number of patients and cycles with dosing delay according to the relationship

Original table:

| Reasons for delays | N | % |
|-----------------------------------|---|------|
| No. of cycles with dosing delays* | | |
| Treatment-related | X | XX.X |
| Hematological | | |
| Non-hematological | | |
| Both | | |
| Non-treatment-related | | |

<sup>(\*)</sup> Denominator= Number of cycles susceptible to have a delay.

**Changed to:** 

| Reasons for | or delays | N | % |
|-------------|-------------------------------------|---|------|
| Cycles | No. of cycles with dosing delays* | | |
| | Treatment-related | X | XX.X |
| | Hematological | | |
| | Non-hematological | | |
| | Both | | |
| | Non-treatment-related | | |
| Patients | No. of patients with dosing delays* | | |
| | Treatment-related | X | XX.X |
| | Hematological | | |
| | Non-hematological | | |
| | Both | | |
| | Non-treatment-related | | |

<sup>(\*)</sup> Denominator= Number of *patient*/cycles susceptible to have a delay.

## Table 12.1.3.2 Number of patients and cycles with dose reduction, any relationship

**Original table:** 

| N | % |
|---|---|
|---|---|

| No. of patients treated | X | XX.X |
|---------------------------------------------------------------|---|------|
| No. of patients with any dose reduced | | |
| No. of patients with: | | |
| No PM01183 reduction | | |
| 1 cycle with PM01183 dose reduced | | |
| 2 cycles with PM01183 dose reduced | | |
| No. of cycles administered | | |
| No. of cycles susceptible to have any dose reduced* | | |
| No. of cycles with PM01183 dose reduced ** | | |
| No. of cycles with PM01183 dose reduced (Treatment-related)** | | |

## **Changed to:**

| | N | % |
|---------------------------------------------------------------|---|------|
| No. of patients treated | X | XX.X |
| No. of patients susceptible to have a dose reduced | | |
| No. of patients with any dose reduced | | |
| No. of patients with: | | |
| No PM01183 reduction | | |
| 1 cycle with PM01183 dose reduced | | |
| 2 cycles with PM01183 dose reduced | | |
| No. of cycles administered | | |
| No. of cycles susceptible to have any dose reduced* | | |
| No. of cycles with PM01183 dose reduced ** | | |
| No. of cycles with PM01183 dose reduced (Treatment-related)** | | |

# Table 12.1.3.3 Number of patients and cycles with dose reduction according to the relationship

#### **Original table:**

| 01.8 | | |
|-------------------------------------|---|------|
| Reasons for reductions | N | % |
| No. of cycles with dose reductions* | | |
| Treatment-related | X | XX.X |
| Hematological | | |
| Non-hematological | | |
| Both | | |
| Non-treatment-related | | |

<sup>(\*)</sup> Denominator= Number of cycles susceptible to have a dose reduction.

#### Changed to:

| Changea to | <b>.</b> | | |
|----------------|---------------------------------------|---|------|
| Reasons for re | eductions | N | % |
| Cycles | No. of cycles with dose reductions* | | |
| | Treatment-related | X | XX.X |
| | Hematological | | |
| | Non-hematological | | |
| | Both | | |
| | Non-treatment-related | | |
| Patients | No. of patients with dose reductions* | | |
| | Treatment-related | X | XX.X |
| | Hematological | | |
| | Non-hematological | | |
| | Both | | |
| | Non-treatment-related | | |

<sup>(\*)</sup> Denominator= Number of *patient*/cycles susceptible to have a dose reduction.

## **Section 12.2.2 Display of Adverse Events**

#### Added:

Table 12.2.2.10 Treatment-related SAEs. Worst grade by patient

| SOC | Preferred Term | Grade<br>1 | | Grade Grade 1 4 | | All* | | |
|---|---|---|---|---|---|---|---|---|
| | | N | % | | N | % | N | % |
| Blood and lymphatic | Anemia NOS | | | | | | | |
| system disorders | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.2.2.11 Treatment-related SAEs. Worst grade by cycle

| SOC | Preferred Term | Grade<br>1 | | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|
| | | N | % | <br>N | % | N | % |
| Blood and lymphatic | Anemia NOS | | | | | | |
| system disorders | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | |

<sup>\*</sup> Any grade

Table 12.2.2.12 SAEs regardless of relationship. Worst grade by patient

| SOC | Preferred Term | Grade<br>1 | | de Grade 4 | | ade<br>4 | All* | |
|---|---|---|---|---|---|---|---|---|
| | | N | % | | N | % | N | % |
| Blood and lymphatic system disorders | Anemia NOS | | | | | | | |
| system disorders | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | |
| Curature disorders | | | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.2.2.13 SAEs regardless of relationship. Worst grade by cycle

| SOC | Preferred Term | Gr | Grade<br>1 | Grade<br>1 | | Grade<br>1 | | Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | N | % | N | % | N | % | | | | |
| Blood and lymphatic system disorders | Anemia NOS | | | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | | | | |

<sup>(\*)</sup> Any grade

## Listing 12.2.2.6 Treatment-related grade 3-4 AEs. Worst grade per patient

**Original Listing:** 

| Patient id. | Cycle | SOC Name | Preferred term | Grade |
|-------------|-------|----------|----------------|-------|

| Patient id. | Cycle | SOC Name | Preferred term | Grade |
|-------------|-------|----------|----------------|-------|

# Listing 12.2.2.8 Adverse Events grade 3-4 regardless of relationship. Worst grade per patient

**Original Listing:** 

| Patient id. | Cycle | SOC Name | Preferred term | Grade |
|-------------|-------|----------|----------------|-------|

Changed to:

| Patient id. | <del>Cycle</del> | SOC Name | Preferred term | Grade |
|-------------|------------------|----------|----------------|-------|

#### **Listing 12.3.1.1 SAEs**

**Original Listing:** 

| <u> </u> | ar Bisang | · • | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Patient id. | Preferred term code | Adverse<br>event<br>reported<br>(verbatim) | Status | Grade | Relationship | Onset date | Resolved date | Action | Serious criteria |

**Changed to:** 

| Patient id. | Preferred term code | Adverse<br>event<br>reported<br>(verbatim) | <del>Status</del> | Grade | Relationship | Onset date | Resolved date | Action | Serious criteria |
|---|---|---|---|---|---|---|---|---|---|

#### **Section 12.4.4 Laboratory Values Over Time**

#### **Tables:**

12.4.4.11 Platelet count time course pattern (summary)

12.4.4.12 Platelet count time course pattern (freqs)

12.4.4.13 Neutrophil count time course pattern (summary)

12.4.4.14 Neutrophil count time course pattern (freqs)

12.4.4.15 AST time course pattern (summary)

12.4.4.16 AST time course pattern (freqs)

12.4.4.17 ALT time course pattern (summary)

#### **Original table headers:**

| | Dose received | | Total |
|---------|---------------|---------|-------|
| 7 mg FD | 6 mg FD | 5 mg FD | Total |

| | Dose received | | |
|----------------------|----------------------|---------------------|-------|
| 7 mg FD / <b>3.5</b> | 6 mg FD / <b>2.6</b> | 5 mg FD/ <b>2.0</b> | Total |
| mg/m <sup>2</sup> | $mg/m^2$ | mg/m <sup>2</sup> | |

## Table added:

Table 11.4.4.18 ALT time course pattern (freqs)

| Table 11.4.4.18 ALT time con | | i Gregs) | Do | se received | | | | |
|---|---|---|---|---|---|---|---|---|
| | 7 mg | FD/3.5 | 6 n | ig FD / 2.6 | 5 1 | ng FD/ 2.0 | | Total |
| | | mg/m²<br>% | N | mg/m² | N | mg/m <sup>2</sup> | N | % |
| Baseline grade 0 | | | | /0 | | /0 | | 70 |
| | | 1 <sup>st</sup> cycle | | | | | | |
| Onset day grade 3/4 | | | | | | | | |
| ≤ 7<br>8-14 | | | | | | | | |
| 6-14<br>≥15 | | | | | | | | |
| ••• | $2^{nd}$ | cycle, 3 <sup>rd</sup> cy | cle | • | | <u> </u> | l | |
| Onset day grade 3/4 | | | | | | | | |
| ≤ <i>7</i> | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| ··· | | Total | | | | | | |
| Onset day grade 3/4 | | 1 Oiul | | | | | | |
| ≤ <i>7</i> | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥15 | | | | | | | | |
| Baseline grade 1, 2 | | | | | | I | | |
| Total | | | | | | | | |
| Total | | 1 <sup>st</sup> cycle | | | | | | |
| Onset day grade 3/4 | | 1 cycle | | | | | | |
| ≤ 7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥15 | | | | | | | | |
| *** | and | cycle, 3 <sup>rd</sup> cy | | | | | | |
| Onset day grade 3/4 | | cycie, 5 ° cy | cie | • | | | | |
| ≤7 | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| ••• | | | | | | | | |
| | | Total | | | | 1 | I | |
| Onset day grade 3/4<br>≤ 7 | | | | | | | | |
| ≥ /<br>8-14 | | | | | | | | |
| ≥ 15 | | | | | | | | |
| Peak day grade 3/4 | | | | | | | | |
| ≤ <i>7</i> | | | | | | | | |
| 8-14 | | | | | | | | |
| ≥ 15<br>Recovery day to grade ≤ 2 | | | | | - | | | |
| Recovery ady to grade ≤ 2<br>≤ 22 | | | | | | | | |
| 23-28 | | | | | | | | |
| ≥ 29 | | | | | L | | <u>L</u> | |
| Duration in days to grade 2 | | | | | | | | |
| ≤5 | | | | | | | | |
| 6-10 | | | | | | | | |
| ≥11 | | | | | | | | |
| Recovery day to grade ≤ 1<br>≤ 22 | | | | | | | | |
| <i>≟ ##</i> | | | 1 | | 1 | l | | |

| | | Dose received | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | 7 n | 7 mg FD / 3.5<br>mg/m <sup>2</sup> | | $ \begin{array}{ccc} 6 \text{ mg } FD/2.6 & 5 \text{ mg } FD/2. \\ \text{mg/m}^2 & \text{mg/m}^2 \end{array} $ | | ng FD/ 2.0<br>mg/m <sup>2</sup> | Total | |
| | N | % | N | % | N | % | N | % |
| 23-28 | | | | | | | | |
| ≥ 29 | | | | | | | | |
| Duration in days to grade 1 | | | | | | | | |
| ≤5 | | | | | | | | |
| 6-10 | | | | | | | | |
| ≥11 | | | | | | | | |

## Listing 12.5.2.3 Troponin I and Troponin T values. Evolution during the study.

**Original listing:** 

| Patient id. | Cycle | Value | ULN |
|-------------|-------|-------|-----|

Changed to:

| Patient id. | Cycle | Test | Value | ULN |
|-------------|-------|------|-------|-----|

# Table 12.6.1 Concomitant medication during treatment (ATC1, ATC2 and ATC4 levels)

**Original table:** 

| Concomitant medication at baseline | N | % |
|------------------------------------|---|---|
| Alimentary tract and metabolism | | |
| Antacids | | |
| Magnesium compounds | | |
| Magnesium adipate | | |
| Blood and blood forming organs | | |
| Antithrombotic agents | | |
| Vitamin K antagonists | | |
| Acenocoumarol | | |

| Changes to: | 2.7 | 0/ |
|------------------------------------|-----|----|
| Concomitant medication at baseline | N | % |
| Alimentary tract and metabolism | | |
| Antacids | | |
| — Magnesium compounds | | |
| Magnesium adipate | | |
| Blood and blood forming organs | | |
| Antithrombotic agents | | |
| - Vitamin K antagonists | | |
| Acenocoumarol | | |

Table 12.6.2 Summary of concomitant medication during treatment

Original table:

| | N | % |
|------------------------------------------|---|---|
| No. of systems at BL (ATC1 level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥3 | | |
| Median (range) | | |
| No. of indications at BL (ATC2 level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥3 | | |
| Median (range) | | |
| No. of agent families at BL (ATC4 level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥3 | | |
| Median (range) | | |
| No. of agents at BL (PN level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥3 | | |
| Median (range) | | |

**Changed to:** 

| Changed to: | | |
|-------------------------------------------------|---|---|
| | N | % |
| No. of systems <i>at BL</i> (ATC1 level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥3 | | |
| Median (range) | | |
| No. of indications <i>at BL</i> (ATC2 level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥3 | | |
| Median (range) | | |
| No. of agent families <i>at BL</i> (ATC4 level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥3 | | |
| Median (range) | | |
| No. of agents at BL (PN level) | | |
| 0 | | |
| 1 | | |
| 2 | | |
| ≥3 | | |
| Median (range) | | |

Table 12.6.5 Transfurions and G-CSF by dose

Table added:

Table 12.6.5 Transfusions and G-CSF by dose

| | 7 mg | g FD | $3.5 \text{ mg/m}^2$ | | Total | |
|--------------|------|------|----------------------|---|-------|---|
| | N | % | N | % | N | % |
| Transfusions | | | | | | |
| RBC | | | | | | |
| Platelets | | | | | | |
| G-CSF | | | | | | |

Rest of tables in this section has been renumbered.

**Section 13 DB Listings** 

**Original title:** 

Listing 13.1.1: Cover

**Changed to:** 

**Listing 13.1.1: Investigator comments** 

Added:

ICH Listings.

- -Listing 16.2.1 Discontinued patients
- -Listing 16.2.2 Protocol deviations
- -Listing 16.2.3 Patients excluded from the efficacy analysis
- -Listing 16.2.4 Demographic data
- -Listing 16.2.5 Compliance and-or Drug Concentration Data
- -Listing 16.2.6 Individual Efficacy Response data
- -Listing 16.2.7 Adverse event listings
- -Listing 16.2.8 Individual laboratory measurements